| Document<br>Type: | Statistical analysis plan |
|---|---|
| Official Title: | Study on the <u>Association</u> of Uterine <u>Perforation</u> and IUD <u>Expulsion</u> With Breastfeeding Status at the Time <u>of IUD</u> Insertion and Postpartum Timing of IUD Insertion in Electronic Medical Record Databases - A Postmarketing Requirement for Mirena (APEX IUD) |
| NCT Number: | NCT03754556 |
| <b>Document Date:</b> | 24 Oct 2018 |



## Statistical analysis plan

| Study on the <u>Association of Uterine Perforation and IUD Expulsion With Breastfeeding Status at</u> the Time of <u>IUD</u> Insertion and Postpartum Timing of IUD Insertion in Electronic Medical Record Databases – A Postmarketing Requirement for Mirena (APEX IUD) | | | |
|---|---|---|---|
| Medicinal product: | Mirena®, Skyla®, Liletta®, Kyleena®, and ParaGard® intrauterine devices | | |
| Study<br>Purpose: | This is a United States postmarketing requirement study assessing outcomes of uterine perforation and intrauterine device (IUD) expulsion in association with breastfeeding, time since delivery, and type of IUD. | | |
| | The study aims to quantify the rist the following comparisons: | study aims to quantify the risk of uterine perforation and IUD expulsion for following comparisons: | |
| | <ul> <li>Women who are breastfeed breastfeeding at the time</li> </ul> | eding at the time of IUD insertion v<br>of IUD insertion | ersus not |
| | <ul> <li>Women who had a first observed IUD insertion within different time<br/>periods postpartum (i.e., ≤ 6 weeks, &gt; 6 weeks and ≤ 14 weeks, &gt; 14 weeks<br/>and ≤ 52 weeks) versus women who had their first observed IUD insertion<br/>more than 52 weeks postpartum, including women without a recorded<br/>delivery within the past 52 weeks</li> </ul> | | |
| | • | nis study will also assess the risk of perforation and expulsion (separately) by pe of IUD. In addition, this study aims to assess the following interactions: | |
| | <ul> <li>The extent to which type of IUD (levonorgestrel-releasing vs. copper IUD) modifies the association between perforation and/or expulsion and breastfeeding status and/or postpartum status</li> </ul> | | |
| | | <ul> <li>The extent to which breastfeeding status modifies the association between<br/>perforation and/or expulsion and postpartum status</li> </ul> | |
| IMPACT<br>No.: | 19682 | Protocol Date: | 29 June 2018 |
| SAP<br>Version,<br>Date: | Version 2.0, 24Oct2018 | SAP includes TLF<br>Specification: | yes 🖂<br>no 🗌 |
| Author: | RTI Health Solutions<br>200 Park Offices Drive<br>Research Triangle Park, NC, US | :A | |



#### Confidential

The information provided in this document is strictly confidential and is intended solely for the guidance of the study. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the study or its use for any other purpose without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) are not displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

This Statistical Analysis Plan is produced on a word-processing system and bears no signatures.

The approval of the Statistical Analysis Plan is documented in a separate signature document.



## **Table of Contents**

| 1 | Introduction | 5 |
|---|---|---|
| 1.1 | Background | |
| 1.2 | Protocol Version and Amendments | 6 |
| 2 | Study Objectives | 6 |
| 2.1 | Primary Objectives | |
| 2.1 | Secondary Objectives | |
| | Study Design | |
| 3.1 | Exposures | |
| 3.2 | Outcomes | |
| 3.3 | Baseline Demographic and Clinical Characteristics | |
| 3.4 | Procedure-Related Characteristics | |
| 3.5 | Indicators of a Difficult IUD Insertion | |
| 3.6 | Provider-Related Characteristics (Not Captured in RI Data) | |
| 3.7 | Start and Stop Dates | |
| 3.8 | Other Parameters | 16 |
| 4 | General Statistical Considerations | 16 |
| 4.1 | General Principles | |
| 4.1.1 | | |
| 4.1.2 | | |
| 4.1.3 | Crude Cumulative Incidence | 17 |
| 4.1.4 | | |
| 4.1.5 | | |
| 4.1.6 | | |
| 4.1.7 | | |
| 4.1.8 | | |
| 4.1.9 | | |
| 4.1.1 | | |
| 4.2 | Handling of Loss to Follow-Up and Premature Discontinuation | |
| 4.3 | Handling of Missing Data | |
| 4.4 | Interim Analyses and Data Monitoring | |
| 4.5 | Data Rules | |
| 4.6 | Definition of Derived Variables and Subgroups | 23 |
| <b>5</b> . | | |
| 5.1 | Analysis Sets | |
| 5.1<br>5.1.1 | | |
| 5.1.1 | | |
| 5.1.2<br>5.1.3 | • | |
| | 2 | |
| | Statistical Methodology | |
| 6.1 | Population Characteristics | |
| 6.2 | Analysis of Primary Variable(s) | |
| 6.2.1 | | |
| 6.2.2 | | |
| 6.3 | Analysis of Secondary Variable(s) | 30 |



| 6.3. | 1 Analysis of IUD Expulsion | 30 |
|---|---|---|
| 6.3. | 2 Analysis of Difficult Insertion | 31 |
| 6.3. | | |
| 6.4 | Safety Analysis | 31 |
| 6.5 | Analysis of Representativeness | |
| 6.6 | Additional Analyses Planned to be Reported Outside the Study Report | 32 |
| 7 | Document History and Changes in the Planned Statistical Analysis | 32 |
| 8 | References | 32 |
| 9 | Appendix | 34 |
| 9.1 | Study Objectives With Corresponding Exposures, Analysis Sets, and Effect E | stimates for |
| | Uterine Perforation | 35 |
| 9.2 | Study Objectives With Corresponding Exposures, Analysis Sets and Effect Es | stimates for |
| | IUD Expulsion | 36 |
| 9.3 | Propensity Score Models Defined by Exposure and Outcomes of Interest | 37 |
| 9.4 | List of Planned Analysis Tables and Figures | 39 |
| 9.5 | Analysis Table Layouts | 43 |
| 9.6 | Illustration of Continuous Enrollment and Look-Back Time for Kaiser Perman | nente Sites |
| | (KPNC, KPSC, and KPWA) | 71 |



#### **Abbreviations**

| BMI | Body Mass Index |
|---|---|
| CI | Confidence Interval |
| EHR | Electronic Health Record |
| EURAS-IUD | European Active Surveillance Study for Intrauterine Devices |
| FDA | Food and Drug Administration |
| ICD-9-CM | International Classification of Diseases, 9th Revision, Clinical Modification |
| ICD-10-CM | International Classification of Diseases, 10th Revision, Clinical Modification |
| IRD | Incidence Rate Difference |
| IRR | Incidence Rate Ratio |
| IUD | Intrauterine Device |
| KPNC | Kaiser Permanente Northern California |
| KPSC | Kaiser Permanente Southern California |
| KPWA | Kaiser Permanente Washington |
| LB | Lower Bound (of the 95% confidence interval) |
| LNG | Levonorgestrel |
| LNG-IUD | Levonorgestrel-Releasing Intrauterine System |
| PMR | Postmarketing Requirement |
| RI | Regenstrief Institute |
| RTI-HS | RTI Health Solutions, a unit of RTI International, a nonprofit research organization |
| SAP | Statistical Analysis Plan |
| TLF | Tables, Listings and Figures |
| TM | Trademark |
| UB | Upper Bound (of the 95% confidence interval) |
| US | United States |

#### 1 Introduction

#### 1.1 Background

Mirena, a levonorgestrel (LNG)-releasing intrauterine system, was approved for use in the United States (US) in December 2000 (Bayer HealthCare Pharmaceuticals Inc., 2015). In August 2015, Bayer received a postmarketing requirement from the US Food and Drug Administration (FDA) to evaluate the incidence of and risk factors for uterine perforation in US women receiving Mirena intrauterine devices (IUDs) at postpartum intervals reflecting US clinical practice (communication from FDA to Bayer, 18 August 2015). Bayer proposed to conduct a retrospective cohort study of women with LNG-IUD or copper IUD in four electronic health record (EHR) databases to assess the risk of uterine perforation and IUD expulsion and potential risk factors, including breastfeeding at the time of IUD insertion, timing of postpartum IUD insertion, and type of IUD (LNG-IUD vs copper). After communication from the FDA in May 2018, Bayer added an assessment of uterine perforation and IUD expulsion by indication for use (as evidenced by diagnosis of heavy menstrual bleeding).



The study aims to quantify the risk of uterine perforation and IUD expulsion for the following comparisons:

- Women who are breastfeeding at the time of IUD insertion versus not breastfeeding at the time of IUD insertion
- Women who had a first observed IUD insertion within different time periods postpartum
   (i.e., ≤ 6 weeks, > 6 weeks and ≤ 14 weeks, > 14 weeks and ≤ 52 weeks) versus women who
   had their first observed IUD insertion more than 52 weeks postpartum, including women
   without a recorded delivery within the past 52 weeks

This study will also assess the risk of perforation and expulsion (separately) by type of IUD. In addition, this study aims to assess the following interactions:

- The extent to which type of IUD (LNG-releasing vs. copper IUD) modifies the association between perforation and/or expulsion and breastfeeding status and/or postpartum status
- The extent to which breastfeeding status modifies the association between perforation and/or expulsion and postpartum status

#### 1.2 Protocol Version and Amendments

Bayer submitted a protocol for the postmarketing requirement (PMR) study to the FDA that was formally accepted for FDA review on 13 December 2017 (PMR #3129-1). On 18 April 2018, the FDA provided comments and recommendations on the protocol that were further clarified in e-mail exchanges between Bayer and the FDA on 23 April and 01 May 2018. The updated protocol (version 2.0) was submitted to the FDA on 29 June 2018 (with this statistical analysis plan) and is aligned to this original version of the statistical analysis plan (version 1.0). The updated protocol (version 2.0) was approved by the FDA (via e-mail) on September 11, 2018.

## 2 Study Objectives

The overall goal of this study is to assess the impact of breastfeeding and timing of postpartum IUD insertion on uterine perforation and IUD expulsion in a population of US women. The study aims to quantify the risk of perforation and expulsion associated with breastfeeding and early postpartum IUD insertion as well as by IUD type and indication for use (e.g., IUD used with concomitant heavy menstrual bleeding). The study includes the following objectives:

#### 2.1 Primary Objectives

- 1. To evaluate whether the risk of uterine perforation among women who were breastfeeding at the time of the first observed IUD insertion differs from the risk of uterine perforation among women who were not breastfeeding at the time of the first observed IUD insertion.
- 2. To evaluate whether the risk of uterine perforation among women who had a first observed IUD insertion within different time periods postpartum (i.e., ≤ 6 weeks, > 6 weeks and ≤ 14 weeks, > 14 weeks and ≤ 52 weeks) differs from the risk of uterine perforation among women who had their first observed IUD insertion more than 52 weeks postpartum, including women without a recorded delivery within the past 52 weeks.



## 2.2 Secondary Objectives

Rates: uterine perforation

- 3. To estimate the incidence rate and cumulative incidence of uterine perforation among women using IUDs
- 4. To estimate the incidence rate and cumulative incidence of uterine perforation among women using IUDs for the following categories of timing of IUD insertion:
  - ≤ 6 weeks postpartum
  - > 6 weeks and  $\leq 14$  weeks postpartum
  - > 14 weeks and  $\le 52$  weeks postpartum
  - > 52 weeks postpartum, including women without recorded delivery within the past
     52 weeks
  - ≤ 14 weeks postpartum
  - > 14 weeks postpartum, including women without recorded delivery within the past
     52 weeks
  - ≤ 36 weeks postpartum
  - > 36 weeks postpartum, including women without recorded delivery within the past
     52 weeks
- 5. To estimate the incidence rate and cumulative incidence of uterine perforation among women who were and were not breastfeeding at the time of IUD insertion
- 6. To estimate the incidence rate and cumulative incidence of uterine perforation among women with different types of IUD (i.e., LNG-IUD and copper IUD)
- To estimate the incidence rate and cumulative incidence of uterine perforation among women with and without menorrhagia (heavy menstrual bleeding) in the 12 months before IUD insertion

Rates: IUD expulsion

- To estimate the incidence rate and cumulative incidence of IUD expulsion among users of IUDs
- 9. To estimate the incidence rate and cumulative incidence of IUD expulsion among users of IUDs for the following categories:
  - ≤ 6 weeks postpartum
  - > 6 weeks and ≤ 14 weeks postpartum
  - > 14 weeks and  $\le 52$  weeks postpartum
  - > 52 weeks postpartum, including women without recorded delivery within the past
     52 weeks
  - ≤ 14 weeks postpartum



- > 14 weeks postpartum, including women without recorded delivery within the past
   52 weeks
- ≤ 36 weeks postpartum
- > 36 weeks postpartum, including women without recorded delivery within the past
   52 weeks
- 10. To estimate the incidence rate and cumulative incidence of IUD expulsion among women who were and were not breastfeeding at the time of IUD insertion
- 11. To estimate the incidence rate and cumulative incidence of IUD expulsion among women with different types of IUD (i.e., LNG-IUD and copper IUD)
- 12. To estimate the incidence rate and cumulative incidence of IUD expulsion among women with and without menorrhagia in the 12 months before IUD insertion

#### Prevalence of difficult IUD insertion

13. To describe the prevalence of indicators of a difficult IUD insertion (e.g., need for cervical dilation or ultrasound guidance, clinician experience) among all users

#### Comparative: uterine perforation

- 14. To estimate the adjusted hazard ratio of uterine perforation among women who had a first observed IUD insertion early in the postpartum period (i.e., ≤ 14 weeks postpartum) versus those who had a first observed IUD insertion late in the postpartum period (i.e., > 14 weeks postpartum, including women without recorded delivery within the past 52 weeks)
- 15. To estimate the adjusted hazard ratio of uterine perforation among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks (this objective will be performed as a sensitivity analysis; same cut point as in EURAS-IUD)
- 16. To estimate the adjusted hazard ratio of uterine perforation for women whose first observed IUD was a copper IUD versus women whose first observed IUD was an LNG-IUD
- 17. To estimate the adjusted incidence rate ratio (IRR) and incidence rate difference (IRD) of uterine perforation at 1 year and 5 years of follow-up among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks (same analytic approach as EURAS-IUD)
- 18. To estimate the adjusted hazard ratios of uterine perforation described in objectives 1, 2, and 14-16 across all subsequent insertions (i.e., not the first insertion) observed within the data. (The site-specific analyses will be performed only if there are more than 20,000 subsequent IUD insertions for that site. The pooled analysis will include all sites regardless of the number of subsequent IUD insertions at a site.)
- 19. To estimate the adjusted hazard ratio of uterine perforation for women using and IUD who have at least one diagnosis code indicating menorrhagia in the 12 months before IUD insertion versus IUD users who do not have this indication (this analysis will be performed



only if more than 20,000 IUD users with an indication of menorrhagia can be included in the analysis)

Comparative: IUD expulsion

- 20. To estimate the adjusted hazard ratio of IUD expulsion among women who were breastfeeding at the time of the first observed IUD insertion versus those who were not breastfeeding at the time of the first observed IUD insertion
- 21. To estimate the adjusted hazard ratio of IUD expulsion for women who had a first observed IUD insertion early in the postpartum period (i.e., ≤ 14 weeks postpartum) versus those who had a first observed IUD insertion late in the postpartum period (i.e., > 14 weeks postpartum, including women without recorded delivery within the past 52 weeks)
- 22. To estimate the adjusted hazard ratio of IUD expulsion for women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery in the past 52 weeks
- 23. To estimate the adjusted hazard ratios of IUD expulsion for women who had a first observed IUD insertion in early postpartum categories versus women who had a first observed IUD insertion late in the postpartum period, using the following strata:
  - ≤ 6 weeks postpartum
  - > 6 weeks and  $\leq 14$  weeks postpartum
  - > 14 weeks and  $\le 52$  weeks postpartum
  - > 52 weeks postpartum, including women without recorded delivery in the past 52 weeks (referent category)
- 24. To estimate the adjusted hazard ratio for IUD expulsion for women whose first observed IUD was an LNG-IUD versus women whose first observed IUD was a copper IUD
- 25. To estimate the adjusted IRR and IRD of IUD expulsion at 1 year and 5 years of follow-up among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks
- 26. To estimate the adjusted hazard ratios of IUD expulsion described in objectives 20-24 across all subsequent insertions (i.e., not the first insertion) observed within the data. (The site-specific analyses will be performed only if there are more than 20,000 subsequent IUD insertions for that site. The pooled analysis will include all sites regardless of the number of subsequent IUD insertions at a site.)
- 27. To estimate the adjusted hazard ratio of IUD expulsion for women using an IUD who have at least one diagnosis code indicating menorrhagia in the 12 months before IUD insertion versus IUD users who do not have this indication (this analysis will be done only if more than 20,000 IUD users with an indication of menorrhagia can be included in the analysis)

Interactions (effect modification)

28. To evaluate the extent to which breastfeeding status (yes vs. no) modifies the association of uterine perforation for women with IUD insertion at different time periods postpartum (i.e., IUD insertion ≤ 14 weeks versus IUD insertion > 14 weeks postpartum) among women



with a recorded delivery within the past 52 weeks at the time of the first observed IUD insertion

- 29. To evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modifies the association between uterine perforation among women who were and were not breastfeeding at the time of the first observed IUD insertion
- 30. To evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modifies the association between IUD expulsion among women who were and were not breastfeeding at the time of the first observed IUD insertion
- 31. To evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modifies the association of uterine perforation for women with IUD insertion at different time periods postpartum (i.e.,  $\leq 6$  weeks, > 6 and  $\leq 14$  weeks, > 14 and  $\leq 52$  weeks) versus IUD insertion more than 52 weeks postpartum, including no recorded delivery within the past 52 weeks at the time of the first observed IUD insertion
- 32. To evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modifies the association of IUD expulsion for women with IUD insertion at different time periods postpartum (i.e.,  $\leq 6$  weeks, > 6 and  $\leq 14$  weeks, > 14 and  $\leq 52$  weeks) versus IUD insertion more than 52 weeks postpartum, including no recorded delivery within the past 52 weeks at the time of the first observed IUD insertion

## 3 Study Design

A retrospective cohort study design will be used to evaluate uterine perforation and IUD expulsion among women who have an IUD insertion identified within EHR data. The study will consider the impact of breastfeeding status at the time of IUD insertion and timing of IUD insertion during the postpartum period on the outcomes of perforation and expulsion.

The earliest possible start for a patient to be eligible for the study population of women with IUD insertion will be 01 January 2001 (after approval of Mirena), and the latest date for a patient to be included in the study population will be 2 months before the end date of the data pull (anticipated to be approximately 30 June 2018 to coincide with anticipated approval of the protocol). The study start date at each study site will be determined by the earlier of (1) the date when Mirena was approved or (2) the date when EHRs were implemented in the four research sites—Kaiser Permanente Northern California (KPNC), Kaiser Permanente Southern California (KPSC), Regenstrief Institute (RI), and Kaiser Permanente Washington (KPWA). Further, the start date at each site for inclusion in the breastfeeding assessment will be dictated by the date at which breastfeeding data became available (Figure 1).



Figure 1. Start and End Dates of EHR Data and Breastfeeding Data, Including First and Last Potential Index Dates, by Data Source

EHR = electronic health records; KPNC = Kaiser Permanente Northern California; KPSC = Kaiser Permanente Southern California; KPWA = Kaiser Permanente Washington; RI = Regenstrief Institute. Note: RI EHRs were implemented prior to 2001.

This study will include all women with evidence of an IUD insertion that have at least 12 months of enrollment history preceding IUD insertion (RI, which does not have enrollment dates, will require a clinical visit at least 12 months before IUD insertion). The first observed IUD insertion for each woman that meets study inclusion/exclusion criteria will be included in the primary analyses. All eligible IUD insertions occurring during the study period will be included in the study for a subset of secondary analysis (objectives 18 and 26).

Each IUD insertion is eligible for inclusion in the study if the database has evidence of insertion of an IUD during the study time window and the woman has been continuously enrolled in the database for at least 12 months before the IUD insertion. IUD insertions will be excluded from the study if a woman is aged more than 50 years at the time of the IUD insertion (IUD insertions that occur in eligible patients at younger ages will be included).

Patients will be followed from the time of IUD insertion until the first occurrence of any of the following: uterine perforation, IUD expulsion, IUD removal, indication of IUD reinsertion, indication of new pregnancy, hysterectomy, death, expiration of IUD, disenrollment from the database, or end of the study period. All person-time at risk that meets these criteria will be included, and there will be no requirement for minimum or maximum follow-up time. All IUD insertions occurring with at least 12 months of enrollment before the insertion that are noted within the data sources will be included in the study. The index date will be captured for each insertion, and baseline data will be collected for each index date (Figure 2). The main analyses for the study will



assess only the first observed IUD insertion for each woman in the database. Secondary analyses will be conducted assessing subsequent insertions (i.e., not the first IUD insertion), as recorded in the database. The sequential number of each insertion, as captured in the data for each woman, will be collected and included as a baseline covariate within these secondary analyses.

At least 12 months
continuous
enrollment

Index Date

Study time

Baseline variables

Outcome variables

Censoring variables

Provider characteristics
Procedure-related characteristics
Indicators of difficult insertion

Figure 2. Covariate data collection around index date

Exposures of postpartum status (based on pregnancy delivery date), breastfeeding status, IUD type, and menorrhagia (as a proxy for indication of use) will be assessed as of the index date of IUD insertion. Outcomes of uterine perforation and IUD expulsion will be assessed beginning on the index date. Baseline data—such as patient demographics, patient characteristics (e.g., personal history of gynecologic conditions such as endometriosis), procedure characteristics, medications, and comorbid conditions (e.g., diabetes)—will be collected from all time in the database before the index date (which will be defined as the day of IUD insertion) and on the index date (Figure 2). Provider characteristics, procedure-related characteristics, and indicators of a difficult insertion will be assessed on the index date (i.e., on the same date or within the same encounter as the index date). The variables to be obtained from each research site are provided in Sections 3.1 through 3.8.

## 3.1 Exposures

- Pregnancy delivery date is the date on which delivery occurred
- Breastfeeding status at the time of IUD insertion: breastfeeding status is defined for every insertion based on whether there is any evidence of breastfeeding (including any breastfeeding or pumping across a 24 hour period) at the time of IUD insertion. For postpartum ≤ 52 weeks, breastfeeding status is defined as Yes, No, or Undetermined. For postpartum > 52 weeks, including no evidence of a live birth in the past 52 weeks, breastfeeding is not assessed (and will be classified as No when used as a covariate).
- IUD type: three-level categorical variable indicating the type of IUD inserted:
  - LNG-IUD: Mirena, Liletta, Skyla, Kyleena
  - Copper IUD: ParaGard, other copper
  - Unknown IUD type



- Menorrhagia: diagnosis of menorrhagia assessed in two variables
  - As an exposure: indicator variable (0 = No, 1 = Yes) for whether the patient was diagnosed with menorrhagia in the year (365 days) prior to or on the index date
  - As a covariate within other exposure assessments: four-level categorical variable for whether the patient was diagnosed with menorrhagia
    - Diagnosed in the year prior to or on the index date, but not diagnosed before that time
    - Not diagnosed in the year prior to or on the index date, but was diagnosed before that time
    - Diagnosis recorded within the year prior to or on the index date and also before that time
    - No diagnosis of menorrhagia within the data

#### 3.2 Outcomes

- Date uterine perforation confirmed is the date on which uterine perforation is documented.
   Either partial or complete perforation will be considered as an outcome, and no distinction will be made between partial and complete perforation.
- Date IUD expulsion confirmed is the date on which IUD expulsion is documented. Either
  partial or complete expulsion will be considered as an outcome, and no distinction will be
  made between partial and complete expulsion.

If both perforation and expulsion occurred on the same date, then the outcome will be classified as both perforation and expulsion, since these outcomes are evaluated separately throughout this study. No analysis will be conducted to assess both perforation and IUD expulsion as a composite outcome or as a subgroup analysis among those with both outcomes.



#### 3.3 Baseline Demographic and Clinical Characteristics

- Age: age in years as of the index date
- Race/ethnicity: categorical variable with nine categories: non-Hispanic white, Hispanic white, non-Hispanic black, Hispanic black, other Hispanic, Asian/Pacific Islander, multiple races/ethnicities, other race/ethnicity, unknown
- Smoking status: indicator variable for smoking status as of the index date (0 = no recent smoking, 1 = recent smoking [active smoker within 365 days prior to or on the index date])
- Body mass index (BMI): continuous variable assessed at the index date or the closest date before or after the index date
- Dysmenorrhea: four-level categorical variable for whether the patient was diagnosed with dysmenorrhea
  - Diagnosed in the year prior to or on the index date, but not diagnosed before that time
  - Not diagnosed in the year prior to or on the index date, but was diagnosed before that time
  - Diagnosis recorded within year prior to or on the index date and also before that time
  - No diagnosis of dysmenorrhea within the data
- Fibroids: indicator variable (0 = No, 1 = Yes) for whether the patient was ever diagnosed with or reported diagnosis of uterine fibroids prior to or on the index date
- Parity: cumulative number of viable pregnancies (i.e., carried to at least 20 weeks gestation)
   prior to and on the index date
- Cesarean delivery will be captured only among women who had at least one delivery prior to the index date and will be captured in two variables:
  - Indicator variable (0 = No, 1 = Yes) for whether the patient *ever had a Cesarean delivery* prior to or on the index date
  - Indicator variable (0 = No, 1 = Yes) for whether the patient had a Cesarean delivery for the most recent delivery that is within 52 weeks prior to or on the index date
- Calendar year of index date: calendar year of the index date (2001-2018, depending on data source)
- Month of index date: calendar month of the index date (1-12 corresponding to January-December, respectively).

#### 3.4 Procedure-Related Characteristics

• The following concomitant gynecological procedures will each be captured as indicator variables (0 = No, 1 = Yes): abortion, aspiration and curettage, dilation and curettage, excision/biopsy of cervix or uterus, ablation, colposcopy and other cervical procedures, hysteroscopy, laminaria, laparoscopy, lysis adhesions, myomectomy, nerve procedure, salpingectomy/oophorectomy. If insufficient data are available to assess (RI only), then concomitant gynecological procedures will be missing.



#### 3.5 Indicators of a Difficult IUD Insertion

- Cervical dilation: indicator variable (0 = No, 1 = Yes) for whether cervical dilation was used during the IUD insertion procedure
- Ultrasound guidance: indicator variable (0 = No, 1 = Yes) for use of ultrasound guidance during placement of the IUD on the day of the IUD insertion
- Paracervical block: indicator variable (0 = No, 1 = Yes) for whether the patient received a
  paracervical block during the IUD insertion procedure
- Provider note indicating a difficult insertion or complicated procedure: indicator variable (0 = No, 1 = Yes) for whether the patient record includes a notation from the provider regarding a difficult insertion or complicated procedure
- Use of misoprostol: indicator variable (0 = No, 1 = Yes) for whether the patient received misoprostol during the 7 days before or on the date of the IUD insertion procedure

## 3.6 Provider-Related Characteristics (Not Captured in RI Data)

- Provider number of IUD insertions in the previous year: number of IUD insertions the provider performed in the previous year as of the index date
- Provider length of employment in the previous year: continuous variable of the number of days employed within the health care system in the past year as of the index date

## 3.7 Start and Stop Dates<sup>1</sup>

- *IUD insertion date* is the date on which IUD insertion is documented
- Beginning date of study period: the first date EHR data are available from the data source for this study (KPNC, KPSC, and KPWA) or the date when Mirena was launched (RI)
- End date of study period: the last date on which EHR data are available from the data source for this study
- Date of start of enrollment (KPNC, KPSC, and KPWA only) is the earliest date of enrollment in the database for the woman (will be used to calculate look-back period)
- Date of first clinical encounter (RI only) is the earliest in-person visit in the database for the woman (will be used to calculate look-back period)
- Date of disenrollment from the database (KPNC, KPSC, and KPWA only) is the date, after the index date, on which the woman was no longer enrolled in an eligible insurance plan (one gap of ≤ 31 days per year will be allowed)
- Date of last clinical encounter in database (RI only) is the last date on which a woman had an in-person encounter that was recorded in the database

<sup>&</sup>lt;sup>1</sup> Note that the actual dates will remain at each data source research partner. The dates may be offset for each patient as an additional data protection measure before transfer of data to RTI-HS.



Censoring date is the earliest of the following dates: date of removal of IUD, date of a
subsequent IUD reinsertion, date of start of new pregnancy, hysterectomy date, date of
bilateral oophorectomy or other type of sterilization, expiration of IUD, death date, date of
disenrollment from database (KPNC, KPSC, and KPWA only) or last clinical encounter (RI
only), and end date of study period

#### 3.8 Other Parameters

- Database: categorical variable of the four data sources included in the study
- Live birth at most recent delivery: indicator variable (0 = No, 1 = Yes) for whether the patient had a pregnancy ending in live birth within the 52 weeks before the index date
- Date of start of most recent (continuous) enrollment (KPNC, KPSC, and KPWA only) is the
  date, prior to the index date, on which the woman started enrollment in an eligible insurance
  plan (one gap of ≤ 31 days per year will be allowed)

#### 4 General Statistical Considerations

All issues concerning patient eligibility, data consistency checks, permissible data modifications, and coding of medical terms and medication will be documented and maintained by research partners following the Data Structure Template (a central document including operational definitions developed by RTI Health Solutions (RTI-HS) and the data source research partners) and the Work Practice Document for quality control. All statistical issues including derived variables are to be detailed in this statistical analysis plan. Determination of sample size was detailed in the study protocol.

#### 4.1 General Principles

The statistical evaluation will be performed by using the software package SAS version 9.4 or higher (SAS Institute Inc., Cary, NC, USA), except when noted otherwise.

The analysis conducted at RTI-HS will follow the relevant RTI-HS standard operating procedures. Programs, logs, and output will be reviewed for accuracy according to the standard operating procedures for programming and quality control. In addition to table creation, some variables will be derived by RTI-HS from the data provided by the research sites; these derived variables are described in Section 4.6. Variables listed in Section 3 will be provided by sites from their databases via use of operational definitions defined by the research team. For data analyses at each site, the standard operating procedures for the site will be used to ensure data quality and security.

#### 4.1.1 Descriptive Analyses

Descriptive analysis of the data will be performed using summary statistics for categorical and quantitative (continuous) data. Continuous data will be described by the number of nonmissing values, median, mean, standard deviation, minimum, and maximum, as well as lower and upper quartiles. Frequency tables will be generated for categorical data. Selected continuous variables will be categorized in a clinically meaningful way or by tertiles of the distribution.



#### 4.1.2 Crude Incidence Rates

Crude incidence rates (I) will be calculated as the number of incident outcomes (E) occurring during the person-time at risk divided by the total person-years at risk (Y).

$$I = \frac{E}{Y}$$

The exact confidence intervals (CIs) will be calculated using the relationship between the Poisson distribution and chi-square distribution as described in Dobson et al. (1991). The lower and upper bounds (LB and UB) of the 95% CI will be calculated as follows:

$$I_{LB} = max\left(0, \left(\frac{X_{2E,0.025}^2}{2}\right)/Y\right), I_{UB} = \left(\frac{X_{2(E+1),0.975}^2}{2}\right)/Y$$

where  $X_{d,a}^2$  represents the ath percentile of the chi-square distribution with d degree of freedom.

Crude incidence rates will be reported as point estimates (number of cases per 1,000 person-years) and 95% CIs.

#### 4.1.3 Crude Cumulative Incidence

Crude estimates of the cumulative incidence, defined as the number of incident outcomes occurring up to a time point out of the number of IUD insertions, will be estimated using the Kaplan-Meier method.

#### 4.1.4 Crude Hazard Ratios

Crude hazard ratios will be estimated using Cox regression models. These crude hazard ratios will be calculated for each outcome without adjustment for covariates. All crude hazard ratios will be reported as point estimates with 95% CIs.

The proportional hazards assumption between each exposure-outcome pairing will be assessed using visual examination of hazard functions, log-log survival curves, and goodness-of-fit testing using Schoenfeld residuals (Kleinbaum and Klein, 2012). Parallel hazard function and log-log survival curves for exposure groups (i.e., the vertical distance between exposure groups is constant) would indicate that the assumption of proportional hazards is met. The hazard function and log-log plot will be generated using the PLOTS=(H LLS) option in the PROC LIFETEST procedure in SAS. The goodness-of-fit global correlation test based on Schoenfeld residuals will be conducted using the ZPH(GLOBAL) option in the PROC PHREG procedure in SAS. A test with P < 0.05 will indicate that the proportional hazards assumption does not hold. If both visual examination and the global correlation test suggest nonproportional hazards, the time-dependent exposure covariate will be included in crude and adjusted hazard ratio models by fitting interaction terms with continuous or categorical time (Paul, 1995). The form of the interaction terms will be determined after reviewing the plots of hazard functions and log-log survival curves. An example SAS program code follows, where *brstime* is the time-dependent exposure covariate created with the programming statement in the PHREG procedure as an exposure-by-time interaction:



```
PROC PHREG DATA=start;

CLASS brstfeed;

MODEL personyr * outcome (0) = brstfeed brstime / TIES=EFRON;

brstime = brstfeed * (personyr > 0.5); /* use 0.5 as an example*/

RUN;
```

For any models including time-dependent exposure covariates, separate hazard ratios will be reported for estimates of the effect of the exposure over time.

#### 4.1.5 Confounder or Bias Adjusted Analyses

Confounding will be controlled through the use of propensity scores, based on the values of covariates at the time of IUD insertion. The propensity score estimates the probability that a given patient will be exposed conditional on measured covariates and can serve as a summary confounder variable. Propensity scores can perform better than conventional regression methods when the number of events relative to the number of potential confounders is small, because rather than having to model the events with many variables, which may lead to overfitting of the outcome model, one can instead model the exposure, for which the larger number of exposed people provides sufficient data to accommodate a rich model (Cepeda et al., 2003). This advantage may be important in this study, given the low number of expected events, particularly for uterine perforation, within this study.

The steps in estimating adjusted exposure effects are listed as follows:

- 1. Derive variables that will be considered for inclusion in the propensity score models.
- 2. Assess balance between exposure groups in the sample.
- Identify key variables to be included in the propensity score model.
- 4. Estimate propensity scores and assess the overlapping area among all exposure groups.
- 5. Calculate weights, normalize the weights, and examine the normalized weights.
- 6. Assess balance between exposure groups in the weighted sample.
- 7. Add to the propensity score model additional terms (e.g., interaction or higher order terms) of the covariates that do not balance.
- 8. Fit the new propensity score model and estimate the propensity scores.
- 9. Repeat steps 5-8 until all the key covariates are balanced.
- 10. Estimate the exposure effect that accounted for the confounders via weighting.

Propensity scores for exposure variables will be estimated by fitting a logistic regression model (for dichotomous exposure variables) or a multinomial logistic regression model (for exposure variables with more than two categories). The dependent variable in the propensity score model is exposure status (e.g., women breastfeeding at the time of IUD insertion vs. not breastfeeding at the time of IUD insertion).

Breastfeeding status, postpartum timing, and IUD type will be included within the propensity score model (as independent variables when not the dependent variable). Other covariates will be assessed



for inclusion in propensity score models based on association with the study outcome (Brookhart et al., 2006); thus, analysts will not be blinded to the outcome. Baseline covariates to be considered for inclusion are listed in Sections 3 and 4.6. Categorical variables will be assessed for inclusion based on indicator coding of the categories. Continuous variables (including integer count variables) will be assessed for inclusion as continuous, dichotomous, and categorical (i.e., indicator coded) variables, as appropriate. Covariates will be included in the propensity score model if the crude hazard ratio is greater than 1.11 or less than 0.90. Additional confounders will be selected for inclusion within propensity score models if at least a 10% change in the hazard ratio of the exposure-outcome relationship occurs when adjusting for that variable, including at least a 10% change in any level of a categorical exposure variable relative to the referent group (> 52 weeks postpartum for postpartum period).

From the fitted logistic regression models, propensity scores and the overlap weights (Li et al., 2018) will be estimated for each IUD insertion. Overlap weighting is a relatively new weighting scheme to adjust for confounding effects. Overlap weights belong to a class of balancing weights, including commonly used weights for inverse probability weighting. Li et al. (2018) mathematically proved and verified in simulations that the overlap weights minimize asymptotic variance among balancing weights. Other advantages of overlap weights over inverse probability weighting include perfect balance for means and bounded weights avoiding explosive weights or the need for arbitrary truncation. In addition, the overlap weights focus on the naturally comparable "overlap" population, and therefore propensity score 'trimming' for a common support area is not necessary. The overlap weights have been applied in observational studies, for example, Schneider et al. (2001), although the term "overlap weights" was not established at that time.

For dichotomous exposure variables, the propensity score is the probability of being exposed. The propensity score for patient (insertion) i is denoted as  $e_i = \Pr(Z_i = 1 | X_i)$ , where  $Z_i$  denotes the exposure (1= exposed, 0 = unexposed), and  $X_i$  denotes a vector of baseline covariates. The overlap weight for patient i is defined as follows:

$$w_i = \begin{cases} 1 - e_i, Z_i = 1 \\ e_i, & Z_i = 0 \end{cases}$$

For categorical exposure variables with more than two levels, the propensity scores will be estimated for each patient and exposure level. Consider an exposure variable with K exposure groups (K > 2). The propensity score for patient i and exposure k, k=1,...K, denoted as  $e_{ik}$ , is the probability that a patient will be exposed to exposure k conditional on measured covariates  $X_i$ :

$$e_{ik} = \Pr(Z_i = k | X_i)$$
, with  $\sum_{k=1}^{K} e_{ik} = 1$ 

The overlap weight for patient *i* given exposure *k* is defined as follows:

$$w_{ik} = \frac{1}{e_{ik} \sum_{k=1}^{K} \frac{1}{e_{ik}}}$$

The overlap weights will be normalized by multiplying the weights by  $\frac{n}{\sum_{i=1}^{n} w_i}$ , where n is the total sample size. The extreme weights (min, max), mean, and standard deviation of the normalized weights will be assessed, although extreme weights are not expected to be an issue with overlap weights because the overlap weights are bounded.



The distribution of propensity scores among exposed (e.g., breastfeeding at the time of IUD insertion) and unexposed (e.g., not breastfeeding at time of IUD insertion) patients will be examined using histograms with kernel smoothing to identify the overlapping area. However, all patients will be included in the analysis when applying overlap weights. The overlap weights put the strong focus on those patients with the highest overlap in their propensity scores and therefore avoid the need for trimming the population.

The balance across exposure groups will be assessed before and after weighting. The distribution of each variable will be compared between categories of the exposure variable, and balance parameters (i.e., standardized differences) (Austin and Stuart, 2015) will be calculated. Pairwise balance parameters (e.g., pairwise standardized differences) will be used for the categorical exposure variable in which each category will be compared to the referent group (> 52 weeks postpartum for postpartum period). The maximum of the pairwise standardized differences will also be reported. The balance between exposure groups will be assessed overall and within each data source. If the groups are unbalanced on key covariates after application of overlap weighting, then the logistic regression model will be revised by including interaction terms (e.g., with data source), higher order terms, or transformation of variables, and the covariate balance between the groups overall and within each data source will be re-evaluated based on the revised model. When satisfactory balance between the exposed and unexposed groups is achieved, the weighting will be incorporated in modeling for confounder-adjusted outcome assessments (Section 4.1.5). The exposure groups are considered balanced if the standardized difference is less than 0.20 (generally considered small) (McCaffrey et al., 2013). If satisfactory balance is difficult to achieve, which is not expected for overlap weighting, matching of patients between groups may be considered.

Separate propensity score models will be developed for exposure-outcome pairings related to breastfeeding status, postpartum period, IUD type, and menorrhagia for uterine perforation and IUD expulsion. The list of propensity score models is provided in Section 9.3. Sections 6.2 and 6.3 includes additional information for specific objectives. In general, the selection of covariates for inclusion in propensity score models will be conducted only using first insertions. The association between baseline covariates and outcomes (crude hazard ratio) will be assessed only using the complete study population, which includes only the first IUD insertion for each woman. No covariate selection will be conducted for *subsequent* insertion models. Instead, for each specific pairing, covariates and terms included in the final propensity score model for first insertions will be included in the propensity score model for subsequent insertions. Additionally, IUD insertion count (the sequential number) may be included in the propensity score model if it is not balanced across exposure groups for *subsequent* insertions. Propensity scores and weights will be estimated from the corresponding propensity score models.

#### 4.1.6 Adjusted Hazard Ratios

The adjusted hazard ratios and 95% CIs will be estimated using weighted Cox regression models. Hazard ratios will be adjusted for possible confounding effects using overlap weighting (Section 4.1.5). This will be conducted in SAS using PROC PHREG with the WEIGHT statement. Normalized weights will be used for the weighted Cox models. The normalized weights add up to the sample size, so that the estimated covariance matrix of the parameter estimators is invariant to the scale of the weights. To account for the fact that the weights are estimated, a robust, sandwichtype variance estimator will be used to calculate 95% CIs. This will be conducted by using the COVSANDWICH option in the PROC PHREG procedure in SAS. Adjusted hazard ratios will be reported as point estimates with 95% CIs.



Time-dependent exposure covariates will be included if violation of the proportional hazards assumption is identified in the unweighted Cox model (described in Section 4.1.4.).

#### 4.1.7 Crude IRR

The crude IRR will be calculated as the crude incidence rate in the exposed divided by the crude incidence rate in the unexposed.

$$IRR = \frac{Incidence\ rate\ in\ the\ exposed}{Incidence\ rate\ in\ the\ unexposed} = \frac{E_1/Y_1}{E_2/Y_2}$$

where  $E_I$  is the number of incident outcomes occurring during person-years at risk in the exposed group,  $Y_I$  is the total person-years at risk in the exposed group,  $E_2$  is the number of incident outcomes occurring during the person-years at risk in the unexposed group, and  $Y_2$  is the total person-years at risk in the unexposed group.

The 95% CI of the crude IRR will be calculated using a Poisson distribution and test-based methods defined in Sahai and Khurshid (1996). The lower and upper bounds of the 95% CI will be calculated as follows:

$$IRR_{LB} = \left(\frac{Y_2}{Y_1}\right) \left(\frac{E_1}{E_2 + 1}\right) \frac{1}{F_{0.025, 2(E_2 + 1), 2E_1}}, IRR_{UB} = \left(\frac{Y_2}{Y_1}\right) \left(\frac{E_1 + 1}{E_2}\right) F_{0.025, 2(E_1 + 1), 2E_2}$$

where  $F_{0.025, vl, v2}$  represents the 2.5th percentile of the F distribution with v1 and v2 degrees of freedom.

All crude IRRs will be reported as point estimates with 95% CIs.

#### 4.1.8 Adjusted IRR Via Weighting

The IRR will be adjusted for possible confounding effects via weighted estimation of the rates using overlap weights (Section 4.1.5) derived from the same propensity score models as those developed for adjustment of the hazard ratios. The adjusted IRR will be calculated as the weighted incidence rate in the exposed divided by the weighted incidence rate in the unexposed.

$$IRR_w = \frac{Weighted incidence \ rate \ in \ the \ exposed}{Weighted incidence \ rate \ in \ the \ unexposed} = \frac{E_{w1}/Y_{w1}}{E_{w2}/Y_{w2}}$$

where  $E_{wl}$  is the number of weighted incident outcomes occurring during person-years at risk in the exposed group,  $Y_{wl}$  is the total weighted person-years at risk in the exposed group,  $E_{w2}$  is the number of weighted incident outcomes occurring during the person-years at risk in the unexposed group, and  $Y_{w2}$  is the total weighted person-years at risk in the unexposed group.

The 95% CI of IRR<sub>w</sub> will be calculated as described in Section 4.1.7 using a Poisson distribution and the number of weighted incident outcomes and weighted person-years.

#### 4.1.9 Crude IRD

The crude IRD will be calculated as the crude incidence rate in the exposed minus the crude incidence rate in the unexposed:

$$IRD = \frac{E_1}{Y_1} - \frac{E_2}{Y_2}$$



with an approximate 95% CI as outlined in Rothman et al. (2008):

$$IRD \pm Z_{0.025} \sqrt{\frac{E_1}{Y_1^2} + \frac{E_2}{Y_2^2}}$$

Where  $Z_{0.025}$  is the 2.5th percentile of the standard normal distribution.

All crude IRDs will be reported as point estimates with 95% CIs.

#### 4.1.10 Adjusted IRD Via Weighting

The IRD will be adjusted for possible confounding effects via weighted estimation of the rates using overlap weights (Section 4.1.5) derived from the same propensity score models as those developed for adjustment of the hazard ratios. The adjusted IRD will be calculated as the weighted incidence rate in the exposed minus the weighted incidence rate in the unexposed.

$$IRD_{w} = \frac{E_{w1}}{Y_{w1}} - \frac{E_{w2}}{Y_{w2}}$$

The 95% CI of IRD<sub>w</sub> will be calculated as described in Section 4.1.9 using the number of weighted incident outcomes and weighted person-years.

#### 4.2 Handling of Loss to Follow-Up and Premature Discontinuation

This is a retrospective study. To minimize use of records with incomplete data for baseline covariates, women will be required to have 12 months of continuous enrollment within the data source prior to the index date. Additionally, at the Kaiser Permanente sites, censoring will occur if more than 31 days passes without insurance coverage sufficient to maintain enrollment.

This study will be conducted using data from four health care systems with EHRs: KPNC, KPSC, KPWA, and RI. Date of disenrollment from the database, that is, the date on which a woman is no longer enrolled in an eligible insurance plan, will be captured by KPNC, KPSC, and KPWA. For RI, date of last clinical encounter—the last date on which a woman has an in-person encounter that is recorded in the database—will be captured. The dates of disenrollment and last clinical encounter will be used as stopping dates for person-time at risk.

#### 4.3 Handling of Missing Data

Missing data will be treated as missing, unless specified otherwise, and no imputations will be performed. In database analyses of previously collected data, if information on a particular binary variable, such as a disease diagnosis or a medication, is available in the database, patients are assumed to have the factor only if there is evidence for its presence (i.e., absence of information will be taken to mean absence of the condition or medication).

Where appropriate, variables will include a "missing" category for analyses. Consequently, data analyses will be conducted using all women and insertions to the extent possible with respect to their observed available data (i.e., the IUD insertion will not be included in an analysis if missing data for any variable in that analysis, except where "missing" is a separate category for the analysis).

Counts of missingness will be reported in descriptive analysis of categorical variables, and percentages for the nonmissing categories will be based on the number of nonmissing values. For continuous variables, the number of nonmissing values will be reported, and descriptive summaries



will be based on the number of nonmissing values. In addition, the percentage of patients or insertions with missing data will be provided for breastfeeding and IUD type.

#### 4.4 Interim Analyses and Data Monitoring

No interim analyses are planned. Data monitoring is not applicable in this retrospective cohort study based on secondary use of EHR data.

#### 4.5 Data Rules

The index date will be the date of the IUD insertion. In the primary analyses, only the first eligible IUD insertion will be considered; all subsequent IUD insertions will be included in secondary analyses (objectives 18 and 26). Baseline characteristics will be assessed for each eligible insertion. The look-back time will consist of all available data on or before the index date, unless otherwise specified for a particular variable in Section 4.6. Because all insertions included in the study are required to have at least 12 months of data before the index date, a minimum of 12 months of data from which to evaluate baseline characteristic values will be available. For some insertions, more information will be available, and all information within the database on or prior to the index date will be considered to reduce misclassification of baseline information.

## 4.6 Definition of Derived Variables and Subgroups

The variables described in Table 1 will be derived by RTI-HS using the data provided by the four research sites. Since the unit of observation in the data provided by the research partners will be an IUD insertion, these variables will be calculated for each insertion and included in the final dataset. If a woman has more than one eligible insertion in the dataset, the variables will be derived for each insertion using data relevant to that insertion.



**Table 1. Definition of Derived Variables** 

| Variable | Definition <sup>a</sup> |
|---|---|
| Baseline covariates | |
| IUD insertion count | The number of eligible IUD insertions for the woman as of the index date (including the index insertion). <i>IUD insertion count</i> increases by 1 each time a new <i>index date</i> is identified for the woman |
| Initial IUD insertion | Indicator variable: If IUD insertion count = 1 then initial IUD insertion = 1 If IUD insertion count > 1 then initial IUD insertion = 0 |
| Difficult insertion | Indicator variable: 1 = Yes if any of the following occur on the index date (or in 7 days before index date for misoprostol): cervical dilation, ultrasound guidance, paracervical block, provider note, use of misoprostol 0 = No if none of the above indicators of difficult insertion are found on the index date |
| Age tertile | Categorical variable for age based on tertiles (or closest integer cut point [i.e., in years]) for all ages at all first index dates observed within the data |
| Duration of look-back period | Derived number of days, starting on the date of start of enrollment or first clinical encounter in the EHR database and ending on the index date Duration of look-back period is calculated for each index date |
| Categorical indicator for<br>provider number of<br>insertions in previous year | Indicator variable: 0 = fewer than 50 provider number of IUD insertions in the 365 days prior to and on the index date, 1 = 50 or more provider number of IUD insertions in the 365 days prior to and on the index date |
| Provider annualized number of insertions in previous year | Provider number of IUD insertions in previous year divided by provider length of employment in previous year, multiplied by 365 |
| Concomitant gynecological procedure | Indicator variable: 1 = Yes if any of the following procedures occurred on the index date: abortion, aspiration and curettage, dilation and curettage, excision/biopsy of cervix or uterus, ablation, colposcopy and other cervical procedures, hysteroscopy, laminaria, laparoscopy, lysis adhesions, myomectomy, nerve procedure, salpingectomy/oophorectomy 0 = No if none of the above procedures occurred on the index date |
| Exposures | |
| Postpartum number of days | Number of person-days, starting on the most recent <i>pregnancy delivery date</i> prior to or on the index date and ending on the <i>index date</i> . There will be a derived <i>postpartum number of days</i> associated with each insertion for each woman. This variable will range from 0 to 365 days and will be missing if the most recent <i>pregnancy delivery date</i> is not recorded or is more than 365 days before the <i>index date</i> . |
| Postpartum—14-week, dichotomous | Indicator variable: * If postpartum number of days ≤ 98, then postpartum—14-week, dichotomous = 1 * If postpartum number of days > 98 or missing, then postpartum—14-week, dichotomous = 0 |



| Variable | Definition <sup>a</sup> |
|---|---|
| Postpartum—36-week, dichotomous | Indicator variable: * If postpartum number of days ≤ 252, then postpartum—36-week, dichotomous = 1 |
| | * If postpartum number of days > 252 or missing, then postpartum—36-week, dichotomous = 0 |
| Postpartum—categorical | Categorical variable: * If postpartum number of days ≤ 42, then postpartum—categorical = 1 (6 weeks or less) * If postpartum number of days > 42 and ≤ 98, then postpartum— categorical = 2 (> 6 to ≤ 14 weeks) * If postpartum number of days > 98 and ≤ 365, then postpartum— categorical = 3 (> 14 to ≤ 52 weeks) |
| | * If postpartum number of days > 365 or missing, then postpartum— categorical = 0 (> 52 weeks or no delivery) |
| Outcomes | |
| Person-time at risk (days, i.e., time to event/censor) | Number of person-days, starting on the <i>index date</i> of IUD insertion and ending on the earliest of <i>date uterine perforation confirmed</i> , <i>date IUD expulsion confirmed</i> , or <i>censoring date</i> . A derived number for <i>person-time at risk</i> will be associated with <b>each</b> <i>IUD insertion</i> for each woman. |
| Uterine perforation event indicator | Indicator variable: 0 = No date of uterine perforation confirmed during the person-time at risk 1 = Yes, date of uterine perforation confirmed during the person-time at risk |
| IUD expulsion event indicator | Indicator variable: 0 = No date of IUD expulsion confirmed during the person-time at risk 1 = Yes, date of IUD expulsion confirmed during the person-time at risk |
| Other parameter | |
| Continuous enrollment | For KPNC, KPSC, and KPWA: Number of days from the latest of beginning date of the study period or date of start of most recent enrollment before the index date to the earliest of end date of study period or date of most recent disenrollment following the index date. See illustration in Section 9.6. For RI: Number of days from the latest of beginning date of the study period or date of first clinical encounter to the earliest of end date of study period or date of last clinical encounter following the index date. |

EHR = electronic health record; IUD = intrauterine device.

## 5 Analysis Sets

## 5.1 Assignment of Analysis Sets

The complete study population will be defined by the study inclusion and exclusion criteria. However, subsets of the complete study population will be used to address certain study objectives. The analysis sets for the *first eligible IUD insertions* are outlined in Table 2. The analysis sets for subsequent IUD insertions will be defined in the same way for the corresponding IUD insertions.

<sup>&</sup>lt;sup>a</sup> Variables in *Italic*, if not defined in this table, are defined in Sections 3.1-3.8.



Table 2. Women Included in Analysis Sets 1 and/or 2

| Event in Electronic Health | Bootportum Status | Breastfeeding Status <sup>a</sup> | | |
|---|---|---|---|---|
| Record | Postpartum Status | Yes | No | Undetermined |
| Delivery in the past year (52 | ≤ 6 weeks | 1, 2 | 1, 2 | 1 |
| weeks) | > 6 weeks and ≤ 14 weeks | 1, 2 | 1, 2 | 1 |
| | > 14 and ≤ 52 weeks | 1, 2 | 1, 2 | 1 |
| No evidence of delivery in the past year | No delivery in the past 52 weeks | NA | 1 | NA |

NA = not applicable.

#### 5.1.1 Analysis Set 1: Complete Study Population

This analysis set will include women with eligible insertions based on study inclusion and exclusion criteria outlined in Section 3 and in the study protocol. This analysis set will include women with missing data for breastfeeding status and/or IUD type for the insertion. The missing data within breastfeeding status and IUD type may be considered a separate group in the analyses (e.g., when developing the propensity score model for postpartum period).

#### 5.1.2 Analysis Set 2: Breastfeeding Status Available

Women who were less than 52 weeks postpartum at the time of IUD insertion and have either "yes" or "no" breastfeeding status at the time of IUD insertion will be included in this analysis set.

Women who have undetermined breastfeeding status for the insertion will not be included.

#### 5.1.3 Analysis Set 3: IUD Type Available

Women with a known type of IUD (either LNG-IUD or copper IUD) for the insertion will be included in this analysis set. Women who have an undetermined IUD type for the insertion will not be included.

## 6 Statistical Methodology

All analyses will be conducted and/or presented using the pooled data and by data source, as appropriate. However, due to the expected sparse outcomes and the data source restriction on reporting IUD type, some analyses will be conducted using only the pooled data, not by data source. In addition, if sparse cells (i.e., count < 10 for exposures, covariates, or outcomes) are identified during the analysis, the sparse cells may be combined into other meaningful categories, excluded from analysis, or left as they are. Decisions will be made by the study team at the time sparse cells are identified.

Objectives and the corresponding exposures, outcomes, analysis sets, and insertions (e.g., first insertions or subsequent insertions) are summarized in Sections 9.1 and 9.2. Propensity score models and the corresponding objectives are summarized in Section 9.3. A list of tables and figures is included in Section 9.4. Table shells are provided as a separate document and are embedded in Section 9.5.

## 6.1 Population Characteristics

Descriptive analyses will be conducted to describe baseline demographics and clinical characteristics at the time of the IUD insertion among the three analysis sets (Analysis Tables 0.1.1 through 0.6.5). Separate tables will be generated for the pooled study population and for each of the

<sup>&</sup>lt;sup>a</sup> The numbers indicate the analysis set numbers.



four databases. Characteristics will be presented overall and for each outcome category of the two study endpoints, perforation and expulsion.

Important characteristics that will be summarized are as follows:

- Demographics (age at index date, race/ethnicity)
- Clinical characteristics (BMI, dysmenorrhea, parity, previous cesarean delivery)
- Procedure-related characteristics (indicator for concomitant procedure and indicators for a difficult IUD insertion [cervical dilation, ultrasound guidance])
- Provider-related characteristics (number of IUD insertions performed)

All variables to be included in the descriptive analyses are described in Sections 3 and 4.6 and listed in the table shells in Section 9.5. Categorical variables will be summarized using frequencies and percentages, and continuous variables will be summarized using means, standard deviations, medians, lower quartiles, upper quartiles, and minimum and maximum values, as described in Section 4.1.1.

Analysis Tables 0.1.1 through 0.3.5 will present demographic summaries for the primary analysis population, which includes only the first observed IUD insertion. Because a woman can have only one eligible insertion in the primary analyses, Analysis Tables 0.1.1 through 0.3.5 will be at the patient level. Analysis Tables 0.4.1 through 0.6.5 will present demographic summaries at the insertion level for the secondary analysis population, which includes all subsequent IUD insertions. Because the unit of observation in the secondary analyses is an IUD insertion, if a woman has more than one eligible insertion during the study period, she will be included more than once in the columns of Analysis Tables 0.4.1 through 0.6.5, with baseline demographic characteristics summarized at each index date. These tables will include number of patients or insertions, as well as number of person-years at risk.

#### 6.2 Analysis of Primary Variable(s)

The primary endpoint in the study is time to diagnosis of uterine perforation (defined in Table 1). Study objectives related to uterine perforation and the corresponding exposures and analysis sets are summarized in Section 9.1. A list of planned analysis tables and figures is included in Section 9.4.

#### 6.2.1 Analysis for Primary Objectives

In the following groups of women, the adjusted hazard ratios for uterine perforation will be evaluated:

- Objective 1. Women who were breastfeeding at the time of the first observed IUD insertion versus those who were not breastfeeding at the time of the first observed IUD insertion.
- Objective 2. Women who had a first observed IUD insertion within different time periods postpartum (i.e., ≤ 6 weeks, > 6 weeks and ≤ 14 weeks, > 14 weeks and ≤ 52 weeks) versus those who had a first observed IUD insertion late in the postpartum period (more than 52 weeks postpartum, including those without recorded delivery in the past 52 weeks).

For objective 1, analyses will be conducted using Analysis Set 2 (breastfeeding status is available). For objective 2, analyses will be conducted using Analysis Set 1 (complete study population). Both analyses will use only the first observed IUD insertion.



Cox regression models will be used to obtain crude hazard ratios overall and by data source with assessment of the proportional hazards assumption (Section 4.1.4).

Confounding effects will be adjusted using the propensity score weighting method (Section 4.1.5). After developing the propensity score model, calculating the weights, and assessing the balance between exposure groups in the weighted sample, adjusted hazard ratios will be estimated using the weighted Cox regression model as described in Section 4.1.6. Additionally, the interaction effect between the data source and the exposure will be assessed after adjustment for confounding. The interaction will be assessed by including terms for exposure, database, and the interaction between the database and the exposure in the weighted Cox models. A type 3 group test for the interaction terms will be conducted. If the test is statistically significant (P < 0.05), then the interaction terms will be retained in the final model, and the adjusted hazard ratios will be reported for each data source. If the interaction terms are not statistically significant, then the interaction terms will be removed, and the overall adjusted hazard ratios (the main effect) will be reported as the results of the primary analyses.

Two-sided 95% CIs of the adjusted hazard ratios for uterine perforation will be presented overall or by data source, as appropriate. If the exposure-by-data source interaction is not significant, then the corresponding two-sided test of the null hypothesis that the natural logarithm of the overall adjusted hazard ratio equals 0 will be performed. The significance level of 0.05 will be applied. There will be no adjustment for multiplicity.

As a sensitivity analysis, confounding effects will be accounted for by including selected key covariates in the unweighted Cox models. The Cox models will include exposure, site, exposure-by-site interaction, and baseline covariates. Due to the sparse outcomes, limited covariates will be selected for inclusion based on their association with the study outcome. The sensitivity analysis will be conducted only for the primary objectives.

Planned Analysis Tables 1.1 (for breastfeeding status) and 2.1 (for postpartum status) will present crude hazard ratio and hazard ratio adjusted via overlap weighting. Analysis Tables 1.2.1 through 1.3.5 and 2.2.1 through 2.3.5 will present baseline characteristics by exposure and standardized differences (described in Section 4.1.5) prior to and after overlap weighting. Analysis Tables 1.4 and 2.4 will present hazard ratios adjusted by including baseline covariates in the model. Results related to the development of propensity score models will be presented in Analysis Tables 33.1.1, 33.2.1, 33.2.2, 33.3.1, 33.3.2 and Analysis Figures 33.1.1 and 33.1.2.

#### 6.2.2 Analysis for Secondary Objectives

#### 6.2.2.1 Crude Incidence Rates and Cumulative Incidence

Crude incidence rates during follow-up and crude cumulative incidence at year 1 and year 5 for the first observed IUD insertions will be calculated overall and by exposure groups (objectives 3-7, as described in Sections 4.1.2 and 4.1.3). Analyses will be conducted using the pooled data and by data source (Analysis Tables 3.1 through 5). Due to data source restrictions, any results on type of IUD by data source will not be reported.

Additionally, the cumulative incidence curve over time, also known as the failure function (i.e., 1 - survival function), will be estimated using the Kaplan-Meier method and plotted overall for each analysis set (Analysis Figures 3.1 through 7.1).



#### 6.2.2.2 Comparing Adjusted Hazard Ratios Among First Observed IUD Insertions

Adjusted hazard ratios associated with the first observed IUD insertions will be estimated for secondary objectives 14-16, and 19 using the same analysis approach (i.e., overlap weighting) as described in Section 6.2.1, with the following exceptions.

- 1. For type of IUD, analyses may be conducted by data source. However, due to data source restrictions, any results on type of IUD by data source will not be reported.
- 2. For secondary objectives that include dichotomization of "early" and "late" postpartum categories, separate propensity score models will not be developed. Rather, the propensity score model developed for the four-category variable will be used. The propensity score for dichotomous exposed group will be calculated by collapsing multiple categories (e.g., propensity score for ≤ 14 weeks = propensity score for ≤ 6 weeks + propensity score for > 6 to ≤ 14 weeks).
- 3. The analyses for objective 19 (menorrhagia) will be performed only if more than 20,000 IUD insertions with an indication of menorrhagia can be included in the analysis.

Balance will be assessed between exposure groups prior to and after weighting. Crude hazard ratios will also be reported.

The same set of analysis tables and figures as those created for objective 1 will be generated, except that no sensitivity analyses will be conducted for these secondary objectives.

## 6.2.2.3 Comparing Adjusted IRR and Adjusted IRD

To compare results from this study to those obtained in EURAS-IUD, we will estimate the adjusted IRR and IRD of uterine perforation at 1 year and 5 years of follow-up among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks (objective 17). Adjusted IRRs and IRDs will be calculated via weighted estimation of the rates using overlap weights as described in Sections 4.1.8 and 4.1.10, respectively.

Using the final analysis datasets after propensity score development and weighting, we will calculate adjusted IRRs and IRDs for the study outcomes. Tables will display the weighted number of outcomes, total weighted person-years, and weighted incidence rates for women who had a first observed IUD insertion  $\leq$  36 weeks postpartum and for women who had a first observed IUD insertion > 36 weeks postpartum. The adjusted IRRs and IRDs along with 95% CIs will be displayed. Analysis Tables 17.1 will be created for uterine perforation.

#### 6.2.2.4 Comparing Adjusted Hazard Ratios for Subsequent IUD Insertions

Adjusted hazard ratios associated with subsequent IUD insertions will be estimated for secondary objectives 18. These analyses will be conducted using the same analysis approach (i.e., Cox models with overlap weights) described previously for first insertions except using subsequent IUD insertions.

Propensity score models will be developed using subsequent IUD insertions. IUD insertion count (the sequential number) may be included in the propensity score model, as needed. To account for the correlation within women with multiple IUD insertions, a robust, sandwich-type variance estimator will be used to calculate 95% CIs. This will be conducted by using the COVSANDWICH



option in the PROC PHREG procedure in SAS. This is the same variance estimator to account for the fact that the weights are estimated.

The site-specific analyses will be performed only if there are more than 20,000 subsequent IUD insertions for that site. The pooled analysis will include all sites regardless of the number of subsequent IUD insertions at individual sites. The crude and adjusted hazard ratios and 95% CIs will be reported.

#### 6.2.2.5 Assessing Effect Modification

Estimation of effect modification of the adjusted hazard ratios will be conducted for secondary objectives 28, 29, 31. The crude and adjusted hazard ratios will be estimated as described in Sections 4.1.4 and 4.1.6 within each level of the potential effect modifier. Due to the expected sparse outcomes and the data source restriction on IUD type, these analysis will be conducted only using the pooled data, not by data source.

For objective 28, the Cox model will include breastfeeding status, early ( $\leq$  14 weeks) versus late (> 14 weeks) postpartum status, and their interaction. The *P* value of the type 3 group test for interaction will be reported. The hazard ratio for breastfeeding status (yes vs. no) will be reported within each level of early ( $\leq$  14 weeks) and late (> 14 weeks) postpartum status. The hazard ratio for postpartum status ( $\leq$  14 weeks vs. > 14 weeks) will be reported within each level of breastfeeding status. In addition, for reporting purposes, the group of no breastfeeding and > 14 weeks postpartum will be considered the referent, and hazard ratios will be reported for postpartum period  $\leq$  14 weeks and breastfeeding,  $\leq$  14 weeks and no breastfeeding, and > 14 weeks and breastfeeding. The adjusted hazard ratio will be obtained using the weighted Cox model. One propensity score model using these four (2 x 2) categories as the dependent variable will be developed. Balance on baseline covariates among the four categories in the weighted sample will be assessed.

For objectives 29 and 31, the Cox models will include the exposure of interest (breastfeeding status or postpartum categories), IUD type, and the interaction between exposure and IUD type. The *P* value of the type 3 group test for interaction will be reported. The hazard ratio for the exposure of interest will be reported within each level of IUD type. The adjusted hazard ratio will be obtained using the weighted Cox model. The weights will be estimated using the same propensity score models developed for the exposure-outcome pairing (Section 9.3).

#### 6.3 Analysis of Secondary Variable(s)

#### 6.3.1 Analysis of IUD Expulsion

The secondary endpoint in the study is time to diagnosis of IUD expulsion (defined in Table 1). In the following groups of women, the adjusted hazard ratios for IUD expulsion will be evaluated:

- Objective 20. Women who were breastfeeding at the time of the first observed IUD insertion versus those who were not breastfeeding at the time of the first observed IUD insertion.
- Objective 23. Women who had a first observed IUD insertion within different time periods postpartum (i.e., ≤ 6 weeks, > 6 weeks and ≤ 14 weeks, > 14 weeks and ≤ 52 weeks) versus those who had a first observed IUD insertion late in the postpartum period (more than 52 weeks postpartum, including those without recorded delivery in the previous 52 weeks).

Study objectives related to IUD expulsion and the corresponding exposures and analysis sets are summarized in Section 9.2 Analyses will be the same as those for uterine preformation, as described



in Section 6.2, except (1) no sensitivity analyses will be conducted and (2) assessment of effect modification using a Cox model including breastfeeding status, early ( $\leq$  14 weeks) versus late (> 14 weeks) postpartum status, and their interaction will not be conducted.

#### 6.3.2 Analysis of Difficult Insertion

The prevalence of indicators of a difficult insertion (objective 13) will be presented via contingency tables including frequencies and percentages of each level of each exposure and outcome variable for five individual indicators of difficult IUD insertion—cervical dilation, ultrasound guidance, paracervical block, provider note, use of misoprostol—plus an indicator for *any* difficult insertion. Analyses will be conducted for the first observed IUD insertion using the pooled data and by data source (Analysis Tables 13.1-13.5). In addition, difficult insertion indicators will be included in summary tables of baseline characteristics.

## 6.3.3 Impact of Transition From ICD-9-CM to ICD-10-CM<sup>2</sup>

The results of this study are dependent on accurate capture of data from source files based on definitions of variables in this study. Since variables will be determined from diagnosis codes (ICD-9-CM, ICD-10-CM), Current Procedural Terminology codes, medication codes (National Drug Codes), and clinical notes (e.g., via natural language processing software) there is a possibility of misclassification. Algorithms for the outcome variables (uterine perforation and IUD expulsion) have been validated in these four databases prior to use of ICD-10-CM coding. No formal validation of the algorithms with ICD-10-CM codes to identify uterine perforation or IUD expulsion will be performed. However, the rate of these outcomes will be reviewed before and after implementation of ICD-10-CM coding to ensure consistency over time. Specifically, 01 October 2015 is the date of transition from ICD-9-CM to ICD-10-CM. The "before" time period will be defined as 01 October 2014 through 30 September 2015, and the "after" time period will be defined as 01 October 2015 through 30 September 2016. The number of patients with an outcome in each time period and the number of patients enrolled in each time period will be reported by data source research partners. The percentage of patients with an outcome among enrolled patients in each time period will be calculated. This analysis will be conducted using the "complete study population" defined in Section 5.1. The count and percentage will be reported for each outcome before and after the transition in the pooled data and by data source (planned Analysis Table 34.1).

## 6.4 Safety Analysis

No additional safety analysis is planned.

## 6.5 Analysis of Representativeness

The study will include all eligible patients identified from KPNC, KPSC, KPWA, and RI. This will cover the following geographic regions in the United States: northern California, southern California, Washington, and Indiana. Summary statistics for demographics and other baseline characteristics of the study cohorts will be provided as described in Section 6.1.

<sup>&</sup>lt;sup>2</sup> ICD-9-CM = International Classification of Diseases, 9th Revision, Clinical Modification; ICD-10-CM = International Classification of Diseases, 10th Revision, Clinical Modification.



# 6.6 Additional Analyses Planned to be Reported Outside the Study Report No additional analyses are planned.

## 7 Document History and Changes in the Planned Statistical Analysis

- Final statistical analysis plan (SAP) v1.0, dated 29 June 2018 initial version, submitted to FDA.
- SAP v2.0, dated 24 October 2018
  - The methods for confounder- or bias-adjusted analyses (previously Section 6.5) was moved to Section 4.1.5 as requested by FDA.
  - Section 4.1.5 (previously Section 6.5) was updated to state that a covariate will be included in the propensity score model if there is "at least a 10% change" rather than "a 10% change."
  - Section 4.1.5 (previously Section 6.5) was revised to include key potential
    confounders (breastfeeding status, postpartum timing, and IUD type) within the
    propensity score model (as independent variables when not the dependent
    variable). Changes were also made to Section 4.1.6 (previously Section 4.1.5) and
    6.2.2.3 to incorporate this change. Section 4.1.8 and 4.1.11 were removed as they
    were no longer needed.
  - The name of the baseline covariate "colposcopy" was changed to "colposcopy and other cervical procedures."

#### 8 References

- Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Stat Med. 2015 Dec 10;34(28):3661-79.
- Bayer HealthCare Pharmaceuticals Inc. Mirena (levonorgestrel-releasing intrauterine system) [prescribing information]. October 2015. Available at: <a href="http://www.accessdata.fda.gov/drugsatfda\_docs/label/2015/021225s031lbl.pdf">http://www.accessdata.fda.gov/drugsatfda\_docs/label/2015/021225s031lbl.pdf</a>. Accessed October 14, 2016.
- Brookhart MA, Schneeweiss S, Rothman KJ, Glynn RJ, Avorn J, Sturmer T. Variable selection for propensity score models. Am J Epidemiol. 2006 Jun 15;163(12):1149-56.
- Cepeda MS, Boston R, Farrar JT, Strom BL. Comparison of logistic regression versus propensity score when the number of events is low and there are multiple confounders. Am J Epidemiol. 2003 Aug 1;158(3):280-7.
- Dobson AJ, Kuulasmaa K, Eberle E, Scherer J. Confidence intervals for weighted sums of Poisson parameters. Stat Med. 1991 Mar;10(3):457-62.
- Kleinbaum DG, Klein M. Evaluating the proportional hazards assumption. In: Kleinbaum DG, Klein M, editors. Survival analysis: a self-learning text, 3rd edition. New York: Springer-Verlag; 2012. p. 161-200.



- Li F, Morgan KL, Zaslavsky AM. Balancing covariates via propensity score weighting. J Am Stat Assoc. 2018 2018/01/02;113(521):390-400.
- McCaffrey DF, Griffin BA, Almirall D, Slaughter ME, Ramchand R, Burgette LF. A tutorial on propensity score estimation for multiple treatments using generalized boosted models. Stat Med. 2013 Aug 30;32(19):3388-414.
- Paul AD. Interactions with time as time-dependent covariates. In: Survival analysis using the SAS® system: a practical guide. Cary, NC: SAS Institute, Inc.; 1995.
- Rothman KJ, Greenland S, Lash TL, editors. Modern epidemiology. 3rd ed. Philadelphia: Lippincott Williams & Wilkins; 2008.
- Sahai H, Khurshid A. Statistics in epidemiology: methods, techniques, and applications.. Boca Raton, FL: CRC Press LLC; 1996.
- Schneider EC, Cleary PD, Zaslavsky AM, Epstein AM. Racial disparity in influenza vaccination: does managed care narrow the gap between African Americans and whites? JAMA. 2001 Sep 26;286(12):1455-60.



## 9 Appendix



## 9.1 Study Objectives With Corresponding Exposures, Analysis Sets, and Effect Estimates for Uterine Perforation

| | Objectives (Identified by Number) and Effect Estimates Related to Uterine Perforation | | | | ed to Uterine |
|---|---|---|---|---|---|
| Exposure<br>(Analysis Set) | Crude IR,<br>cum.<br>incidence<br>(first<br>insertion) | Adj. HR via<br>weighting,<br>crude HR<br>(first<br>insertion) | Adj. HR via<br>weighting,<br>crude HR<br>(subsequent<br>insertions) | Weighted IRR<br>and IRD (at 1 year<br>and 5 years),<br>crude IRR and<br>IRD<br>(first insertion) | Adj. and crude<br>HR within each<br>level of the<br>modifier (first<br>insertion) |
| Breastfeeding<br>(AS2) | 5 | 1ª | 18 | | 28, interaction with ≤ 14 vs > 14 weeks postpartum 29, modified by IUD type |
| 4-level<br>postpartum<br>(AS1) | 4 | 2ª | 18 | | 31, modified by<br>IUD type |
| ≤ 14 wks vs. > 14<br>weeks<br>postpartum<br>(AS1) | 4 | 14 | 18 | | |
| ≤ 36 wks vs. > 36<br>weeks<br>postpartum<br>(AS1) | 4 | 15 | 18 | 17 | |
| IUD type <sup>b</sup> (AS3) | 6 | 16 | 18 | | |
| Menorrhagia<br>(AS1) | 7 | 19 | | | |
| Overall (AS1,<br>AS2, AS3) | 3 | | | | |

AS1 = Analysis Set 1: complete study population; AS2 = Analysis Set 2: breastfeeding status available; AS3 = Analysis Set 3: IUD type available; HR = hazard ratio; IR = incidence rate; IRD = incidence rate difference; IRR = incidence rate ratio; IUD = intrauterine device.

<sup>&</sup>lt;sup>a</sup> Also, regression adjustment will be conducted as a sensitivity analysis.

<sup>&</sup>lt;sup>b</sup> Aggregated analysis only, not by site.


# 9.2 Study Objectives With Corresponding Exposures, Analysis Sets and Effect Estimates for IUD Expulsion

| | Objectives | Identified by N | lumber) and Effect | Estimates Related to | IUD Expulsion |
|---|---|---|---|---|---|
| Exposure<br>(Analysis Set) | Crude IR,<br>cum.<br>incidence<br>(first<br>insertion) | Adj. HR via<br>weighting,<br>crude HR<br>(first<br>insertion) | Adj. HR via<br>weighting,<br>crude HR<br>(subsequent<br>insertions) | Weighted IRR<br>and IRD (at 1 year<br>and 5 years),<br>crude IRR and<br>IRD<br>(first insertion) | Adj. and crude<br>HR within each<br>level of the<br>modifier (first<br>insertion) |
| Breastfeeding (AS2) | 10 | 20 | 26 | | 30, modified by IUD type |
| 4-level<br>postpartum<br>(AS1) | 9 | 23 | 26 | | 32, modified by<br>IUD type |
| ≤ 14 wks vs. > 14<br>weeks<br>postpartum<br>(AS1) | 9 | 21 | 26 | | |
| ≤ 36 wks vs. > 36<br>weeks<br>postpartum<br>(AS1) | 9 | 22 | 26 | 25 | |
| IUD type <sup>a</sup> (AS3) | 11 | 24 | 26 | | |
| Menorrhagia<br>(AS1) | 12 | 27 | | | |
| Overall (AS1,<br>AS2, AS3) | 8 | | | | |

AS1 = Analysis Set 1: complete study population; AS2 = Analysis Set 2: breastfeeding status available; AS3 = Analysis Set 3: IUD type available; HR = hazard ratio; IR = incidence rate; IRD = incidence rate difference; IRR = incidence rate ratio; IUD = intrauterine device.

<sup>&</sup>lt;sup>a</sup> Aggregated analysis only, not by site.



### 9.3 Propensity Score Models Defined by Exposure and Outcomes of Interest

| Model<br>Number | Exposure<br>(Dependent Variable of<br>Propensity Score Model) | Outcome<br>(Not Included<br>in Propensity<br>Score Model) | IUD<br>Insertion | Covariate<br>Selection | Objective<br>Number |
|---|---|---|---|---|---|
| 1 | Breastfeeding status (yes vs. no) | Uterine<br>perforation | First<br>insertion | Yes | 1 (primary<br>objective)<br>29 |
| 2 | Postpartum insertion (4 categories) | Uterine<br>perforation | First<br>insertion | Yes | 2 (primary<br>objective)<br>14 <sup>a</sup><br>15 <sup>a</sup><br>17 <sup>a</sup><br>31 |
| 3 | IUD type (LNG vs. copper) | Uterine perforation | First insertion | Yes | 16 |
| 4 | Menorrhagia (yes vs. no) | Uterine perforation | First insertion | Yes | 19 |
| 5 | Breastfeeding status (yes vs. no) | IUD expulsion | First insertion | Yes | 20<br>30 |
| 6 | Postpartum insertion (4 categories) | IUD expulsion | First<br>insertion | Yes | 23<br>21 <sup>a</sup><br>22 <sup>a</sup><br>25 <sup>a</sup><br>32 |
| 7 | IUD type (LNG vs. copper) | IUD expulsion | First insertion | Yes | 24 |
| 8 | Menorrhagia (yes vs. no) | IUD expulsion | First insertion | Yes | 27 |
| 9 | Interaction of breastfeeding and early vs. late postpartum (breastfeeding/≤ 14 weeks; breastfeeding/> 14 weeks; no breastfeeding/≤ 14 weeks; no breastfeeding/> 14 weeks [referent]) | Uterine<br>perforation | First<br>insertion | Yes | 28 |
| 10 | Breastfeeding status (yes vs. no) | Uterine perforation | Subsequent insertions | No <sup>b</sup> | 18 |
| 11 | Postpartum insertion (4 categories) | Uterine perforation | Subsequent insertions | No <sup>b</sup> | 18 ª |
| 12 | IUD type (LNG vs. copper) | Uterine perforation | Subsequent insertions | No <sup>b</sup> | 18 |
| 13 | Breastfeeding status | IUD expulsion | Subsequent insertions | No <sup>b</sup> | 26 |
| 14 | Postpartum insertion (4 categories) | IUD expulsion | Subsequent insertions | No <sup>b</sup> | 26 a |
| 15 | IUD type (LNG vs. copper) | IUD expulsion | Subsequent insertions | No <sup>b</sup> | 26 |

IUD = intrauterine device; LNG = levonorgestrel.

Reference Number: RD-OI-0215 Supplement Version: 8



<sup>a</sup> Secondary objectives include dichotomization of "early" and "late" postpartum categories. Separate propensity score models will not be *developed* for these objectives. Rather, the propensity scores calculated with the four-category variable will be used. The propensity scores for dichotomous exposure groups will be calculated by collapsing multiple categories (e.g., propensity score for ≤ 14 weeks = propensity score for ≤ 6 weeks + propensity score for > 6 to ≤ 14 weeks).

b Covariates and terms included in the final propensity score model for first insertions will be included in the propensity score model for subsequent insertions. Additionally, IUD insertion count (the sequential number) may be included in the propensity score model if it is not balanced across exposure groups for subsequent insertions.



### 9.4 List of Planned Analysis Tables and Figures

| Table/Figure<br>Number | Content | Table<br>Layout <sup>a</sup> | Note |
|---|---|---|---|
| Population<br>Characteristics | | | |
| Tables 0.1.1<br>through 0.1.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; complete patient population, first insertions | Layout 1 | Pooled and by site (5 tables) |
| Tables 0.2.1<br>through 0.2.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; breastfeeding status available, first insertions | Layout 1 | Pooled and by site (5 tables) |
| Tables 0.3.1<br>through 0.3.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; IUD type available, first insertions | Layout 1 | Pooled and by site (5 tables) |
| Tables 0.4.1<br>through 0.4.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; complete patient population, subsequent insertions | Layout 1 | Pooled and by site (5 tables) |
| Tables 0.5.1<br>through 0.5.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; breastfeeding status available, subsequent insertions | Layout 1 | Pooled and by site (5 tables) |
| Tables 0.6.1<br>through 0.6.5 | Baseline characteristics overall, by uterine perforation and by IUD expulsion; IUD type available, subsequent insertions | Layout 1 | Pooled and by site (5 tables) |
| Objective 1 | Breastfeeding and uterine perforation | | |
| Table 1.1 | Crude and adjusted HR for breast feeding status | Layout 2.1 | Pooled and by site (1 table) |
| Tables 1.2.1<br>through 1.2.5 | Baseline characteristics by exposure and absolute standardized difference | Layout 3.1 | Pooled and by site (5 tables) |
| Tables 1.3.1<br>through 1.3.5 | Baseline characteristics and absolute standardized differences after overlap weighting | Layout 3.1 | Pooled and by site (5 tables) |
| Figure 1.1.1<br>through 1.1.5 | Standardized differences in the unweighted and weighted samples | | Pooled and by site (5 figures) |
| Table 1.4 | Adjusted HR from Cox model with baseline covariates (sensitivity analysis) | Layout 7 | Pooled, including interaction with site (1 table <sup>b</sup> ) |
| Objective 2 | Postpartum period and uterine perforation | | |
| Tables 2.1 | Crude and adjusted HR for postpartum status | Layout 2.2 | Pooled and by site (1 table) |
| Tables 2.2.1<br>through 2.2.5 | Baseline characteristics by exposure and absolute standardized difference | Layout 3.2 | Pooled and by site (5 tables) |
| Tables 2.3.1<br>through 2.3.5 | Baseline characteristics and absolute standardized differences after overlap weighting | Layout 3.2 | Pooled and by site (5 tables) |



| Table/Figure<br>Number | Content | Table<br>Layout <sup>a</sup> | Note |
|---|---|---|---|
| Figure 2.1.1<br>through 2.1.5 | Standardized differences in the unweighted and weighted samples | | Pooled and by site (5 figures) |
| Table 2.4 | Adjusted HR from Cox model with baseline covariates (sensitivity analysis) | Layout 7 | Pooled, including interaction with site (1 table <sup>b</sup> ) |
| Objectives 3 through 12 | Crude incidence rate and cumulative incidence by analysis set, postpartum status, breastfeeding status, IUD type, menorrhagia | | |
| Tables 3.1<br>through 3.5 | Crude incidence rate and cumulative incidence | Layout 8 | Pooled and by site (5 tables) |
| Figure 3.1 | Kaplan-Meier cumulative incidence plot by analysis set | | Pooled (1 figure) |
| Figure 4.1 | Kaplan-Meier cumulative incidence plot by postpartum status | | Pooled (1 figure) |
| Figure 5.1 | Kaplan-Meier cumulative incidence plot by breastfeeding status | | Pooled (1 figure) |
| Figure 6.1 | Kaplan-Meier cumulative incidence plot by IUD type | | Pooled (1 figure) |
| Figure 7.1 | Kaplan-Meier cumulative incidence plot by menorrhagia | | Pooled (1 figure) |
| Objectives 8<br>through 12 | Crude incidence rates and cumulative incidence for IUD expulsion | | Same set of tables and figures as objectives 3-7 (5 tables + 5 figures) |
| Objective 13 | | | |
| Table 13.1<br>through 13.5 | Prevalence of difficult IUD insertion by exposure and outcome | Layout 9 | Pooled and by site (5 tables) |
| Objective 14 | Postpartum period (≤ 14 vs. > 14 weeks) and uterine perforation | | Same set of tables and figures as objective 1 excluding Table 1.4 (11 tables + 5 figures) |
| Objective 15 | Postpartum period (≤ 36 vs. > 36 weeks) and uterine perforation | | Same set of tables and figures as objective 1 excluding Table 1.4 (11 tables + 5 figures) |
| Objective 16 | IUD type and uterine perforation | | Same set of tables and figures as objective 1 excluding Table 1.4 Only pooled results will be reported (3 tables + 1 figures) |
| Objective 17 | Postpartum period (≤ 36 vs. > 36 weeks) and uterine perforation | | |
| Table 17.1 | Crude and adjusted incidence rate ratios and differences for uterine perforation at 1 year and 5 years of follow-up | Layout 10 | Pooled and by site (1 table) |
| Objective 18 <sup>c</sup> | Subsequent insertions for uterine perforation (subsequent insertions) | | Same set of tables and figures as objectives 1, 2, 14, 15, 16 excluding Tables 1.4 and 2.4 (47tables + 21 figures) |
| Objective 19 <sup>d</sup> | Menorrhagia and uterine perforation | | Same set of tables and figures as objective 1 excluding Table 1.4 (11 tables + 5 figures) |



| Table/Figure<br>Number | Content | Table<br>Layout <sup>a</sup> | Note |
|---|---|---|---|
| Objectives 20<br>through 27 <sup>c,d</sup> | Comparative analysis for IUD expulsion | | Same set of tables and figures as objectives 1, 2, 14-19, excluding Tables 1.4 and 2.4 (106 tables + 47 figures) |
| Objective 28 | Effect modification | | |
| Table 28.1 | Effect modification of breastfeeding status and postpartum status on uterine perforation | Layout 11 | Pooled (1 table) |
| Objective 29 | Effect modification | | |
| Table 29.1 | Effect modification of IUD type on breast feeding status and uterine perforation | Layout 12.1 | Pooled (1 table) |
| Objective 30 | Effect modification | | |
| Table 30.1 | Effect modification of IUD type on breast feeding status and IUD expulsion | Layout 12.1 | Pooled (1 table) |
| Objective 31 | Effect modification | | |
| Table 31.1 | Effect modification of IUD type on postpartum status and uterine perforation | Layout 12.2 | Pooled (1 table) |
| Objective 32 | Effect modification | | |
| Table 32.1 | Effect modification of IUD type on postpartum status and IUD expulsion | Layout 12.2 | Pooled (1 table) |
| Development of<br>propensity<br>score models | | | |
| Tables 33.1.1<br>through 33.1.2 | Assessing relationship with outcome: crude HR for baseline covariates | Layout 4 | Pooled (2 tables) |
| Tables 33.2.1<br>through 33.2.9 | Assessing confounding effect: HR adjusted for one covariate | Layout 5 | Pooled (9 tables) |
| Tables 33.3.1<br>through 33.3.15 | Propensity score model | Layout 6 | Pooled (15 tables) |
| Figure 33.1.1<br>through 33.1.15 | Histograms with kernel smoothing of propensity scores by exposure | | Pooled (15 figures) |
| Impact of<br>transition from<br>ICD-9-CM to<br>ICD-10-CM | | | |
| Tables 34.1 | Percentage of uterine perforation or IUD expulsion prior to and after implementation of ICD-10-CM coding | Layout 13 | Pooled and by site (1 table) |

HR = hazard ratio; ICD-9-CM = International Classification of Diseases, 9th Revision, Clinical Modification; ICD-10,CM = International Classification of Diseases, 10th Revision, Clinical Modification; IUD = intrauterine device.

Note: In the report, analysis tables related to IUD type will report only the results across all sites, not by site. However, by-site analyses may be conducted for internal purposes and will not be shared with Bayer.

<sup>&</sup>lt;sup>a</sup> Table layouts are included in Section 9.5.

Reference Number: RD-OI-0215 Supplement Version: 8



- b If breastfeeding status, postpartum timing, or IUD type are not included within a propensity score (as independent variables when not the dependent variable), then a separate Cox model also including these variables as covariates will be developed. If this occurs additional tables will be added using Table Layout 7.
- <sup>c</sup> The analyses by site for objectives 18, and 26 will be done only for sites with more than 20,000 subsequent IUD insertions.
- <sup>d</sup> The analyses for objectives 19 and 27 will be done only if more than 20,000 IUD users with an indication of menorrhagia can be included in the analysis.



#### 9.5 Analysis Table Layouts

This section includes planned table layouts for the analysis. In the title section of the table layouts, words in yellow highlight are subject to change depending on specific analysis.

#### **List of Analysis Table Layouts**

- Table Layout 1. Baseline Characteristics Overall, by Uterine Perforation, and by IUD Expulsion;
  Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 2.1. Hazard Ratios of Uterine Perforation for Breastfeeding Status; Analysis Set:
  Breastfeeding Status Available, First IUD Insertion; Database: Pooled and by Site
- Table Layout 2.2. Hazard Ratios of Uterine Perforation for Postpartum Status; Analysis Set:

  Complete Study Population, First IUD Insertion; Database: Pooled and by Site
- Table Layout 3.1. Baseline Characteristics and Absolute Standardized Differences of Baseline Characteristics for Breastfeeding Status; Analysis Set: Breastfeeding Status Available, First IUD Insertion; Database: Pooled
- Table Layout 3.2. Baseline Characteristics and Absolute Standardized Differences of Baseline Characteristics for Postpartum Status; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 4. Crude Hazard Ratio of Uterine Perforation for Baseline Characteristics; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 5. Hazard Ratio of Uterine Perforation for Postpartum Status and Percent Change After Adjustment for a Single Covariate; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 6. Propensity Score Model for Breastfeeding With Outcome Model for Uterine
  Perforation; Analysis Set: Breastfeeding Status Available, First IUD Insertion; Database:
  Pooled
- Table Layout 7. Adjusted Hazard Ratio of Uterine Perforation for Postpartum Status From Cox Model With Baseline Covariates (Sensitivity Analysis); Analysis Set: Complete Study Population, First IUD Insertion
- Table Layout 8. Crude Incidence Rates and Cumulative Incidence for Uterine Perforation; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 9. Prevalence of Difficult IUD Insertion by Exposure Group and Outcome; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled
- Table Layout 10. Crude and Adjusted<sup>a</sup> Incidence Rate Ratios and Incidence Rate Differences<sup>b</sup> for Uterine Perforation at 1 Year and 5 Years of Follow-up, Comparing Women With a First Observed IUD Insertion ≤ 36 Weeks Postpartum Versus > 36 Weeks Postpartum; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled and by Site
- Table Layout 11. Effect Modification of Breastfeeding Status and Postpartum Status on Uterine Perforation; Analysis Set: Breastfeeding Status Available, First IUD Insertion; Database: Pooled
- Table Layout 12.1. Effect Modification of IUD Type on Breastfeeding Status and Uterine

  Perforation; Analysis Set: Breastfeeding Status Available, First IUD Insertion; Database:
  Pooled
- Table Layout 12.2. Effect Modification of IUD Type on Postpartum Status and Uterine Perforation; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled

Reference Number: RD-OI-0215 Supplement Version: 8



Table Layout 13. Percentage of Uterine Perforation or IUD Expulsion Before and After Implementation of ICD-10-CM Coding; Analysis Set: Complete Study Population, First IUD Insertion; Database: Pooled and by Site

Reference Number: RD-OI-0215

Supplement Version: 8



Table Layout 1. Baseline Characteristics Overall, by Uterine Perforation, and by IUD Expulsion;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled

| | Overall | l | Jterine Perforatio | n | | IUD Expulsion | |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined (N = XX,XXX) |
| Person-years at risk | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X |
| Demographic characteristics | | | | | | | |
| Age, in years | | | | | | | |
| Category <sup>a</sup> , n (%) | | | | | | | |
| Category 1 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Category 2 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Category 3 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Race/ethnicity, n (%) | | | | | | | |
| Asian/Pacific Islander | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Hispanic black | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Hispanic other | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Hispanic white | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Multiple | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Non-Hispanic white | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Non-Hispanic black | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Other | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Unknown | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Recent smoker c, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |



| | Overall | l | Jterine Perforatio | n | IUD Expulsion | | |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Duration of look-back period, in months | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Calendar year of index date, n (%) | | | | | | | |
| 2001 - 20XX | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 20XX - 2018 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Calendar month of index date, n (%) | | | | | | | |
| January | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| December | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Clinical characteristics | | | | | | | |
| BMI, in kg/m <sup>2</sup> | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Dysmenorrhea diagnosis, n (%) | | | | | | | |
| Recent, on or within1 year before the index date only | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Past, more than 1 year before the index date only | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Records in recent and past periods | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| No record of diagnosis | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |



| | Overall | Į | Jterine Perforatio | n | | IUD Expulsion | |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Fibroids, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Parity | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Cesarean delivery before the index dated, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Cesarean delivery for most recent delivery before the index date <sup>d</sup> , n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Procedure-related characteristics | | | | | | | |
| Concomitant gynecological procedure, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Abortion procedure, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Aspiration and curettage, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Dilation and curettage, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Excision/biopsy of cervix or uterus, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Ablation, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Colposcopy and other cervical procedures, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Hysteroscopy procedure, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Laminaria procedure, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Laparoscopy, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Lysis adhesions, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Myomectomy, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Nerve procedure, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Salpingectomy/ oophorectomy, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |



| | Overall | Uterine Perforation IUD Exp | | | | IUD Expulsion | oulsion |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Insertion-related characteristics | | | | | | | |
| IUD insertion count | | | | | | | |
| 1 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 2 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 3 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| continue to other categories | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Any difficult insertion, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Cervical dilation, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Ultrasound guidance, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Paracervical block, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Difficult insertion noted, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Use of misoprostol, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Provider-related characteristics <sup>e</sup> | | | | | | | |
| Number of IUD insertions performed | | | | | | | |
| < 50 insertions, n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | [XX.X, XX.X] | [XX.X, XX.X] | [XX.X, XX.X] | [XX.X, XX.X] | [xx.x, xx.x] | [XX.X, XX.X] | [XX.X, XX.X] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Annualized number of insertions in previous year | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | xx,xxx | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | XX.X<br>[XX.X, XX.X] | XX.X<br>[XX.X, XX.X] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |



| | Overall | l | Jterine Perforatio | n | | IUD Expulsion | Ision |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Length of employment in previous year, in days | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | xx,xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | XX.X<br>[XX.X, XX.X] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Other parameters | | | | | | | |
| Live birth within the past 52 weeks (most recent delivery), n (%) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Continuous enrollment f (months) | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX | XX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Continuous enrollment on or before index date (months) | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XXX,XXX | XX,XXX | XX,XXX | XXX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X<br>[XX.X, XX.X] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] | xx.x<br>[xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Continuous enrollment on or after index date (months) | | | | | | | |
| N | XXX,XXX | XX,XXX | XX,XXX | XXX,XXX | XX,XXX | XX,XXX | XXX,XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median [Q1, Q3] | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |



| | Overall | l | Jterine Perforatio | n | | IUD Expulsion | |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Site (data source) | | , | , , | , | , | , | |
| KPNC | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| KPSC | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| KPWA | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| RI | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Study exposure groups | | | | | | | |
| Breastfeeding status | | | | | | | |
| Yes | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| No | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Undetermined | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Postpartum status | | | | | | | |
| 6 weeks or less | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| > 6 to ≤ 14 weeks | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| > 14 to ≤ 52 weeks | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| > 52 weeks or no delivery | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| ≤ 14 weeks | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| > 14 weeks or no delivery | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| ≤ 36 weeks | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| > 36 weeks or no delivery | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| IUD type | | | | | | | |
| LNG-IUD | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Copper IUD | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Unknown | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |



| | Overall | Į | Jterine Perforatio | n | IUD Expulsion | | |
|---|---|---|---|---|---|---|---|
| Characteristic | (N = XXX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Undetermined<br>(N = XX,XXX) |
| Menorrhagia in the past year | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Diagnosis recorded only within 1 year | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Diagnosis recorded only before 1 year | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Diagnosis recorded both within and before 1 year | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| No diagnosis | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |

BMI = body mass index; IUD = intrauterine device; LNG-IUD = levonorgestrel-releasing intrauterine system; Q1 = lower quartile (i.e., 25th percentile); Q3 = upper quartile (i.e., 75th percentile); SD = standard deviation.

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1</u>: For tables of first insertions, N is number of patients. For tables of subsequent insertions, N is number of insertions.

Programming note 2: For variables with missing data, number of missing data will be reported.

Programming note 3: IUD insertion count will not be shown for tables using only first insertions because it will be 1 for every patient.

Programming note 4: Site (data source) will be shown only for the pooled table, not for the site tables.

Programming note 5: Results by IUD type will be presented only for the pooled table, not by site.

<sup>&</sup>lt;sup>a</sup> Age categories were based on tertiles of the distribution.

<sup>&</sup>lt;sup>b</sup> Available only in the KPSC database.

<sup>&</sup>lt;sup>c</sup> Available in the KPSC database; partially available in the KPWA and RI databases.

<sup>&</sup>lt;sup>d</sup> Cesarean delivery summarized only among women who had at least one delivery before the index date.

<sup>&</sup>lt;sup>e</sup> Available in the KPNC, KPSC, and KPWA databases.

<sup>&</sup>lt;sup>f</sup> Continuous enrollment is not a baseline covariate. It is included only for summary purposes.



Table Layout 2.1. Hazard Ratios of Uterine Perforation for Breastfeeding Status;

Analysis Set: Breastfeeding Status Available, First IUD Insertion;

Database: Pooled and by Site

| Cito | Breastfeeding | Events | Insertions | Bereen weers | Crude UD (05% CI) | Adjusted | |
|---|---|---|---|---|---|---|---|
| Site | Status | Events | insertions | Person-years | Crude HR (95% CI) | HR (95% CI) | P Value |
| Pooled | Yes | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | No | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPNC | Yes | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | No | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPSC | Yes | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | No | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPWA | Yes | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | No | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| RI | Yes | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | No | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.

Note: Crude HRs were estimated from five Cox models using pooled data or within each site. Adjusted HRs were estimated from two Cox models weighted using overlap weights. The adjusted HRs by site were estimated from the Cox model including exposure, site, and site-by-exposure interaction (type 3 group test for interaction: P = 0.xxxx); the overall adjusted HR (reported only if the interaction is not significant) was estimated from the Cox model including exposure and site.

Note: The P value is from the Cox model for the test of the null hypothesis that the adjusted HR equals one.

Note: The proportional hazards assumption was tested using the global correlation test based on Schoenfeld residuals with the pooled data (P = 0.xxxx).

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1:</u> The pooled adjusted HR and related footnote will be shown only if the interaction term is not statistically significant (P > 0.05).

<u>Programming note 2:</u> If the proportional hazards assumption is violated, time-dependent exposure covariates will be included in Cox models. The table above will be expanded to include separate hazard ratios for the effect of exposure over time.

<u>Programming note 3</u>: For tables that include results by IUD type, only pooled results will be presented, not by site.

Programming note 4: For all tables and notes with P values, note that the P in "P value" is capitalized and in italics, and a space (not a hyphen) follows the P.

Reference Number: RD-OI-0215 Supplement Version: 8



Table Layout 2.2. Hazard Ratios of Uterine Perforation for Postpartum Status; Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled and by Site

| Site | Postpartum Status | F4- | Insertions | Person-years | Course LID (OF9) CIV | Adjusted | a |
|---|---|---|---|---|---|---|---|
| | | atus Events | | | Crude HR (95% CI) | HR (95% CI) | P Value |
| Pooled | 6 weeks or less | xx | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 6 to ≤ 14 weeks | XX | xx | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 14 to ≤ 52 weeks | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 52 weeks or no<br>delivery | XX | xx | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPNC | 6 weeks or less | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 6 to ≤ 14 weeks | xx | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 14 to ≤ 52 weeks | XX | xx | xxx,xxx.x | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 52 weeks or no<br>delivery | XX | xx | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPSC | 6 weeks or less | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 6 to ≤ 14 weeks | XX | xx | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 14 to ≤ 52 weeks | XX | xx | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 52 weeks or no<br>delivery | XX | xx | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |
| KPWA | 6 weeks or less | xx | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 6 to ≤ 14 weeks | XX | XX | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 14 to ≤ 52 weeks | XX | xx | XXX,XXX.X | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 52 weeks or no<br>delivery | XX | xx | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |

Reference Number: RD-OI-0215

Supplement Version: 8



| Site | Doots out on Otation | Evente | Insertions | Person-years | Crudo HB (059/ CI) | Adjusted <sup>a</sup> | |
|---|---|---|---|---|---|---|---|
| | Postpartum Status | Events | | | Crude HR (95% CI) | HR (95% CI) | P Value |
| RI | 6 or less weeks | xx | xx | xxx,xxx.x | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 6 to ≤ 14 weeks | xx | xx | xxx,xxx.x | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 14 to ≤ 52 weeks | xx | xx | xxx,xxx.x | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | 0.XXXX |
| | > 52 weeks or no<br>delivery | XX | XX | XXX,XXX.X | 1.00 (Reference) | 1.00 (Reference) | - |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.

Note: Crude HRs were estimated from five Cox models using pooled data or within each site. Adjusted HRs were estimated from two Cox models weighted using overlap weights: The adjusted HRs by site were estimated from the Cox model including exposure, site, and site-by-exposure interaction (type 3 group test for interaction: P = 0.xxxx); the pooled adjusted HR (reported only if the interaction is not significant) was estimated from the Cox model including exposure and site.

Note: The P value is from the Cox model for the test of the null hypothesis that the adjusted HR equals one.

Note: The proportional hazards assumption was tested using the global correlation test based on Schoenfeld residuals with the pooled data (P = 0.xxxx).

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1</u>: The pooled adjusted HR and related footnote will be shown only if the interaction term is not significant (P > 0.05).

Programming note 2: For tables that include results by IUD type, only pooled results will be presented, not by site.



Table Layout 3.1. Baseline Characteristics and Absolute Standardized Differences of Baseline Characteristics for Breastfeeding Status;

Analysis Set: Breastfeeding Status Available, First IUD Insertion;

Database: Pooled

| | Breastfeed | | |
|---|---|---|---|
| Characteristic | Yes<br>(N = XX,XXX) | No<br>(N = XX,XXX) | Absolute Standardized<br>Difference |
| Age, in years | | | |
| Category, n (%) | | | |
| Category 1 | xx (x.x) | xx (x.x) | XX.X |
| Category 2 | xx (x.x) | xx (x.x) | XX.X |
| Category 3 | xx (x.x) | xx (x.x) | XX.X |
| N | XX | xx | |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | XX.X |
| Median [Q1, Q3] | xx.x [xx.x, xx.x] | xx.x [xx.x, xx.x] | |
| Min, max | XX, XX | xx, xx | |
| Continue for other variables under consideration | | | |

IUD = intrauterine device; Q1 = 25th percentile; Q3 = 75th percentile; SD = standard deviation.

Generated using xxxx.sas on xxxxxxx.

Programming note 1: For tables that include results by IUD type, only pooled results will be presented, not by site.



Table Layout 3.2. Baseline Characteristics and Absolute Standardized Differences of Baseline Characteristics for Postpartum Status;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled

| | | Postpartum Status | | | | Absolute Standardized Difference<br>(vs. > 52 Weeks or No Delivery) | | |
|---|---|---|---|---|---|---|---|---|
| Characteristic | 6 Weeks or<br>less<br>(N = XX) | > 6 to ≤ 14<br>Weeks<br>(N = XX) | > 14 to ≤ 52<br>Weeks<br>(N = XX) | > 52 Weeks<br>or No<br>Delivery<br>(N = XX) | 6 Weeks or<br>Less | > 6 to ≤ 14<br>Weeks | > 14 to ≤ 52<br>Weeks | Maximum<br>Difference |
| Age, in years | | | | | | | | |
| Category, n (%) | | | | | | | | |
| Category 1 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | XX.X | XX.X | XX.X | XX.X |
| Category 2 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | XX.X | XX.X | XX.X | XX.X |
| Category 3 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | XX.X | XX.X | XX.X | XX.X |
| N | XX | XX | XX | XX | | | | |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | XX.X | XX.X | XX.X | XX.X |
| Median [Q1, Q3] | xx.x [xx.x,<br>xx.x] | xx.x [xx.x,<br>xx.x] | xx.x [xx.x,<br>xx.x] | xx.x [xx.x,<br>xx.x] | | | | |
| Min, max | XX, XX | XX, XX | XX, XX | XX, XX | | | | |
| Continue for other variables under consideration | | | | | | | | |

IUD = intrauterine device; Q1 = 25th percentile; Q3 = 75th percentile; SD = standard deviation.

<sup>&</sup>lt;sup>a</sup> Age categories were based on tertiles of the distribution.



Table Layout 4. Crude Hazard Ratio of Uterine Perforation for Baseline Characteristics;

Analysis Set: Complete Study Population, First IUD Insertion;

**Database: Pooled** 

| Characteristic | Crude HR (95% CI) |
|--------------------------------------------------|-------------------|
| Age, in years | |
| Category 1 | x.xx (x.xx, x.xx) |
| Category 2 | x.xx (x.xx, x.xx) |
| Category 3 | 1.00 (Reference) |
| Continuous age (scale) | x.xx (x.xx, x.xx) |
| Continue for other variables under consideration | |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.

Note: HRs were estimated from separate Cox models, each of which included only one baseline covariate in the model.

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1:</u> The list of variables maybe adjusted after reviewing the data. This may include rescaling, collapsing levels, or categorizing variables.



Table Layout 5. Hazard Ratio of Uterine Perforation for Postpartum Status and Percent Change After Adjustment for a Single Covariate;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled

| Adjustment Covariate | Postpartum Status | HR (95% CI) | HR % Change<br>After Adjustment | Covariate Included in<br>Final Propensity Score<br>Model |
|---|---|---|---|---|
| No adjustment | 6 weeks or less | x.xx (x.xx, x.xx) | - | |
| | > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) | - | |
| | > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) | - | |
| | > 52 weeks or no delivery | 1.00 (Reference) | | |
| Categorical age | 6 weeks or less | x.xx (x.xx, x.xx) | XX.X | Yes or No |
| | > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) | XX.X | |
| | > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) | XX.X | |
| | > 52 weeks or no delivery | 1.00 (Reference) | | |
| Continuous age | 6 weeks or less | x.xx (x.xx, x.xx) | XX.X | Yes or No |
| | > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) | XX.X | |
| | > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) | XX.X | |
| | > 52 weeks or no delivery | 1.00 (Reference) | | |
| Continue for other variables under consideration | | | | |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1:</u> The list of variables maybe adjusted after reviewing the data. This may include rescaling, collapsing levels, or categorizing variables.



Table Layout 6. Propensity Score Model for Breastfeeding With Outcome Model for Uterine Perforation;

Analysis Set: Breastfeeding Status Available, First IUD Insertion;

**Database: Pooled** 

| Parameter | Coefficient (SE) | P Value |
|---------------------|------------------|---------|
| Intercept | xx | 0.xxxx |
| Covariate 1 | | 0.xxxx |
| Category 1 | xx | - |
| Category 2 | xx | - |
| | xx | - |
| Category reference | Reference | |
| Covariate 2 (scale) | XX | 0.xxxx |

IUD = intrauterine device; SE = standard error.

Note: Postpartum timing and IUD type were included in the propensity score model. Other covariates were included in the propensity score model if the crude hazard ratio was greater than 1.11 or less than 0.90. Additional confounders were selected for inclusion within propensity score models if at least a 10% change in the hazard ratio of the exposure-outcome relationship occurs when adjusting for that variable.



Table Layout 7. Adjusted Hazard Ratio of Uterine Perforation for Postpartum Status From Cox Model With Baseline Covariates (Sensitivity Analysis);

Analysis Set: Complete Study Population, First IUD Insertion

| | Adjusted HR (95% CI) |
|---------------------------|----------------------|
| KPNC | |
| 6 weeks or less | x.xx (x.xx, x.xx) |
| > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) |
| > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) |
| > 52 weeks or no delivery | 1.00 (Reference) |
| KPSC | |
| 6 weeks or less | x.xx (x.xx, x.xx) |
| > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) |
| > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) |
| > 52 weeks or no delivery | 1.00 (Reference) |
| KPWA | |
| 6 weeks or less | x.xx (x.xx, x.xx) |
| > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) |
| > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) |
| > 52 weeks or no delivery | 1.00 (Reference) |
| RI | |
| 6 weeks or less | x.xx (x.xx, x.xx) |
| > 6 to ≤ 14 weeks | x.xx (x.xx, x.xx) |
| > 14 to ≤ 52 weeks | x.xx (x.xx, x.xx) |
| > 52 weeks or no delivery | 1.00 (Reference) |
| Covariate 1 | |
| Category 1 | x.xx (x.xx, x.xx) |
| Category 2 | 1.00 (Reference) |
| Covariate 2 (scale) | x.xx (x.xx, x.xx) |
| Covariate 3 | |
| Category 1 | x.xx (x.xx, x.xx) |
| Category 2 | 1.00 (Reference) |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.



Note: The adjusted HR was estimated from the Cox model including exposure, site, site-by-exposure interaction (type 3 group test for interaction: *P* = 0.xxxx), and listed baseline covariates.

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1:</u> The list of variables will be adjusted after reviewing the data.



Table Layout 8. Crude Incidence Rates and Cumulative Incidence for Uterine Perforation;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled

| Groups | Insertions | Person-years | Events | Crude Incidence<br>Rate <sup>a</sup><br>(95% CI) | 1-Year Crude<br>Cumulative Incidence <sup>b</sup><br>(95% CI) | 5-Year Crude<br>Cumulative Incidence <sup>b</sup><br>(95% CI) |
|---|---|---|---|---|---|---|
| Analysis set | | | | | | |
| Complete study population | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Breastfeeding<br>status available | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| IUD type available | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Postpartum status | | | | | | |
| 6 weeks or less | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| > 6 to ≤ 14 weeks | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| > 14 to ≤ 52 weeks | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| > 52 weeks or no<br>delivery | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| ≤ 14 weeks | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| > 14 weeks or no<br>delivery | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| ≤ 36 weeks | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| > 36 weeks or no<br>delivery | XXX | xxx.x | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Breastfeeding status | | | | | | |
| Yes | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| No | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Undetermined | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| IUD type | | | | | | |
| LNG-IUD | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Copper IUD | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| Unknown | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |

Reference Number: RD-OI-0215

Supplement Version: 8



| Groups | Insertions | Person-years | Events | Crude Incidence<br>Rate <sup>a</sup><br>(95% CI) | 1-Year Crude<br>Cumulative Incidence <sup>b</sup><br>(95% CI) | 5-Year Crude<br>Cumulative Incidence <sup>b</sup><br>(95% CI) |
|---|---|---|---|---|---|---|
| Menorrhagia | | | | | | |
| Yes | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |
| No | XXX | XXX.X | XX | x.xx (x.xx, x.xx) | xx.x% (xx.x%, xx.x%) | xx.x% (xx.x%, xx.x%) |

CI = confidence interval; IUD = intrauterine device; LNG-IUD = levonorgestrel-releasing intrauterine system.

Generated using xxxx.sas on xxxxxxx.

Programming note 1: Summary for IUD type available set and ty IUD type will only be presented in the pooled table, not by site.

<sup>&</sup>lt;sup>a</sup> Incidence rates are expressed per 1,000 person-years.

<sup>&</sup>lt;sup>b</sup> Crude estimate of cumulative incidence, defined as the number of incident outcomes occurring during a specific time period out of the number of IUD insertions during the same time period, were estimated using the Kaplan-Meier method.



Table Layout 9. Prevalence of Difficult IUD Insertion by Exposure Group and Outcome;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled

| Exposure or Outcome Group | | N | Cervical<br>Dilation<br>n (%) | Ultrasound<br>Guidance<br>n (%) | Paracervical<br>Block<br>n (%) | Provider Note n (%) | Use of<br>Misoprostol<br>n (%) | Any<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| All patients | | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Breastfeeding | Yes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Undetermined | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Postpartum status | 6 weeks or less | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 6 to ≤ 14 weeks | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 14 to ≤ 52 weeks | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 52 weeks or no<br>delivery | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IUD type | LNG-IUD | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Copper IUD | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Undetermined | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Menorrhagia | Yes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IUD expulsion | Yes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| - | No | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Uterine perforation | Yes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

IUD = intrauterine device; LNG-IUD = levonorgestrel-releasing intrauterine system.

Generated using xxxx.sas on xxxxxxx.

Programming note 1: Results by IUD type will be presented only for the pooled table, not by site.



Table Layout 10. Crude and Adjusted<sup>a</sup> Incidence Rate Ratios and Incidence Rate Differences<sup>b</sup> for Uterine Perforation at 1 Year and 5 Years of Follow-up, Comparing Women With a First Observed IUD Insertion ≤ 36 Weeks Postpartum Versus > 36 Weeks Postpartum; Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled and by Site

| | | 1 Year of Follow-Up | | 5 Years of Follow-Up | |
|---|---|---|---|---|---|
| Site | | ≤ 36 Weeks | > 36 Weeks or<br>No Delivery | ≤ 36 Weeks | > 36 Weeks or<br>No Delivery |
| Pooled | Events | XX | XX | XX | XX |
| | Person-years | XX.X | XX.X | XX.X | XX.X |
| | Incidence rate | X.XX | X.XX | X.XX | X.XX |
| | Crude IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Crude IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| KPNC | Events | XX | XX | XX | XX |
| | Person-years | XX.X | XX.X | XX.X | XX.X |
| | Incidence rate | X.XX | X.XX | X.XX | X.XX |
| | Crude IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Crude IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| KPSC | Events | XX | XX | XX | XX |
| | Person-years | XX.X | XX.X | XX.X | XX.X |
| | Incidence rate | X.XX | X.XX | X.XX | X.XX |
| | Crude IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Crude IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | | | • | | |



| | | 1 Year of Follow-Up | | 5 Years of Follow-Up | |
|---|---|---|---|---|---|
| Site | | ≤ 36 Weeks | > 36 Weeks or<br>No Delivery | ≤ 36 Weeks | > 36 Weeks or<br>No Delivery |
| KPWA | Events | XX | XX | XX | XX |
| | Person-years | XX.X | XX.X | XX.X | XX.X |
| | Incidence rate | X.XX | X.XX | X.XX | X.XX |
| | Crude IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Crude IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| RI | Events | XX | XX | XX | XX |
| | Person-years | XX.X | XX.X | XX.X | XX.X |
| | Incidence rate | X.XX | X.XX | X.XX | X.XX |
| | Crude IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRR (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Crude IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |
| | Adjusted IRD (95% CI) | x.xx (x.xx, x.xx) | Reference | x.xx (x.xx, x.xx) | Reference |

CI = confidence interval; IRD = incidence rate difference; IRR = incidence rate ratio; IUD = intrauterine device.

Generated using xxxx.sas on xxxxxxx.

<u>Programming note 1</u>: Generate tables x.1 for uterine perforation and x.2 for IUD expulsion.

<sup>&</sup>lt;sup>a</sup> Adjusted via weighted estimation of the rates using overlap weights derived from the same propensity score models as those developed for adjustment of the hazard ratios.

<sup>&</sup>lt;sup>b</sup> Incidence rates and incidence rate differences are expressed per 1,000 person-years.



Table Layout 11. Effect Modification of Breastfeeding Status and Postpartum Status on Uterine Perforation;

Analysis Set: Breastfeeding Status Available, First IUD Insertion;

**Database: Pooled** 

| | | Breastfee | HR (95% CI) | |
|---|---|---|---|---|
| | Postpartum Status | Yes | No | Breastfeeding<br>(Yes vs. No) |
| Number of events/ | 14 weeks or less | xx/xx | xx/xx | |
| insertions | > 14 weeks or no delivery | xx/xx | xx/xx | |
| Crude HR | 14 weeks or less | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 14 weeks or no delivery | x.xx (x.xx, x.xx) | 1.00 (Reference) | x.xx (x.xx, x.xx) |
| | HR (95% CI) 14 weeks or less vs. > 14 weeks or no delivery | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | |
| Adjusted HR | 14 weeks or less | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 14 weeks or no delivery | x.xx (x.xx, x.xx) | 1.00 (Reference) | x.xx (x.xx, x.xx) |
| | HR (95% CI) 14 weeks or less vs. > 14 weeks or no delivery | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | |
| | Type 3 group test for interaction of breastfeeding status and postpartum status | | | P = 0.xxxx |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device.

Note: Crude HRs were estimated from the Cox model including breastfeeding status, postpartum status, and their interaction. Adjusted HRs were estimated from the Cox models including breastfeeding status, postpartum status, and their interaction, weighted using overlap weights.

Reference Number: RD-OI-0215

Supplement Version: 8



Table Layout 12.1. Effect Modification of IUD Type on Breastfeeding Status and Uterine Perforation;

Analysis Set: Breastfeeding Status Available, First IUD Insertion;

**Database: Pooled** 

| Modifier<br>IUD Type | Exposure<br>Breastfeeding Status | Number of<br>Events | Number of<br>Insertions | Crude HR<br>(95% CI) | Adjusted HR<br>(95% CI) |
|---|---|---|---|---|---|
| LNG-IUD | Yes | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | No | XX | XX | 1.00 (Reference) | 1.00 (Reference) |
| Copper IUD | Yes | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | No | XX | XX | 1.00 (Reference) | 1.00 (Reference) |
| Type 3 group test for interaction with breastfeeding status | | | | | P = 0.xxxx |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device; LNG-IUD = levonorgestrel-releasing intrauterine system.

Note: Crude HRs were estimated from the Cox model including breastfeeding status, IUD type, and their interaction. Adjusted HRs were estimated from the Cox models including breastfeeding status, IDU type, and their interaction, weighted using overlap weights.

Supplement Version: 8



Table Layout 12.2. Effect Modification of IUD Type on Postpartum Status and Uterine Perforation;

Analysis Set: Complete Study Population, First IUD Insertion;

**Database: Pooled** 

| Modifier<br>IUD Type | Exposure<br>Postpartum Status | Number of<br>Events | Number of<br>Insertions | Crude HR<br>(95% CI) | Adjusted HR<br>(95% CI) |
|---|---|---|---|---|---|
| LNG-IUD | 6 weeks or less | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 6 to ≤ 14 weeks | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 14 to ≤ 52 weeks | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 52 weeks or no delivery | XX | XX | 1.00 (Reference) | 1.00 (Reference) |
| Copper IUD | 6 weeks or less | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 6 to ≤ 14 weeks | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 14 to ≤ 52 weeks | XX | XX | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| | > 52 weeks or no delivery | XX | XX | 1.00 (Reference) | 1.00 (Reference) |
| Type 3 group test for interaction with postpartum status | | | | | P = 0.xxxx |

CI = confidence interval; HR = hazard ratio; IUD = intrauterine device; LNG-IUD = levonorgestrel-releasing intrauterine system.

Note: Crude HRs were estimated from the Cox model including postpartum status, IUD type, and their interaction. Adjusted HRs were estimated from the Cox models including postpartum status, IDU type, and their interaction, weighted using overlap weights.



Table Layout 13. Percentage of Uterine Perforation or IUD Expulsion Before and After Implementation of ICD-10-CM Coding;

Analysis Set: Complete Study Population, First IUD Insertion;

Database: Pooled and by Site

| | 1-Year Before | | | 1-Year After | | |
|---|---|---|---|---|---|---|
| Site | Patients | Uterine Perforation | IUD Expulsion | Patients | Uterine Perforation | IUD Expulsion |
| | N | n (%) | n (%) | N | n (%) | n (%) |
| Pooled | XX | xx (xx.x) | xx (xx.x) | XX | xx (xx.x) | xx (xx.x) |
| KPNC | XX | xx (xx.x) | xx (xx.x) | XX | xx (xx.x) | xx (xx.x) |
| KPSC | XX | xx (xx.x) | xx (xx.x) | XX | xx (xx.x) | xx (xx.x) |
| KPWA | XX | xx (xx.x) | xx (xx.x) | XX | xx (xx.x) | xx (xx.x) |
| RI | XX | xx (xx.x) | xx (xx.x) | XX | xx (xx.x) | xx (xx.x) |

IUD = intrauterine device.

Generated using xxxx.sas on xxxxxxx.

Programming note 1: Research partners will provide counts for this table.

Reference Number: RD-OI-0215 Supplement Version: 8



## 9.6 Illustration of Continuous Enrollment and Look-Back Time for Kaiser Permanente Sites (KPNC, KPSC, and KPWA)

Scenario 1. One IUD Insertion With No Uterine Perforation or IUD Expulsion



Scenario 2. One IUD Insertion With One Uterine Perforation









Note: if the beginning date of the study period is within the continuous enrollment period (illustrated in the above figures), the beginning date of the study period will be used as the beginning of continuous enrollment. Similarly, if the end date of the study period is within the continuous enrollment period, the end date of the study period will be used as the end of the continuous enrollment.